CLINICAL TRIAL: NCT01667419
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study of Vemurafenib (RO5185426) Adjuvant Therapy in Patients With Surgically Resected, Cutaneous BRAF-Mutant Melanoma at High Risk for Recurrence
Brief Title: A Study of Vemurafenib Adjuvant Therapy in Participants With Surgically Resected Cutaneous BRAF-Mutant Melanoma
Acronym: BRIM8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO27826; 2011-004011-24 (EudraCT Number)
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Cohort 1 Vemurafenib (Experimental): Participants with completely resected Stage IIC, IIIA, or IIIB cutaneous melanoma) received vemurafenib, 960 milligrams (mg) twice daily, in 28-day cycles, for up to 52 weeks
  Interventions: Drug: Vemurafenib
- Cohort 1 Placebo (Placebo Comparator): Participants with completely resected Stage IIC, IIIA, or IIIB cutaneous melanoma) received vemurafenib-matching placebo twice daily, in 28-day cycles, for up to 52 weeks
  Interventions: Drug: Placebo
- Cohort 2 Vemurafenib (Experimental): Participants with Stage IIIC cutaneous melanoma received vemurafenib, 960 mg twice daily, in 28-day cycles, for up to 52 weeks
  Interventions: Drug: Vemurafenib
- Cohort 2 Placebo (Placebo Comparator): Participants with Stage IIIC cutaneous melanoma received vemurafenib-matching placebo twice daily, in 28-day cycles, for up to 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vemurafenib — 4 tablets of vemurafenib 240 mg each (total 960 mg) were administered orally as per the schedule specified in the respective arm.
  Other Names: RO5185426/F17, Zelboraf
  Arms: Cohort 1 Vemurafenib; Cohort 2 Vemurafenib
Drug: Placebo — Placebo matching to vemurafenib were administered orally as per the schedule specified in the respective arm.
  Arms: Cohort 1 Placebo; Cohort 2 Placebo

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled study will evaluate the efficacy and safety of vemurafenib in participants with completely resected, cutaneous BRAF mutation-positive melanoma at high risk for recurrence. Participants will be enrolled in two separate cohorts: Cohort 1 will include participants with completely resected Stage IIC, IIIA (participants with one or more nodal metastasis greater than [>] 1 millimeter [mm] in diameter), or IIIB cutaneous melanoma, as defined by the American Joint Committee on Cancer (AJCC) Classification, Version 7; Cohort 2 will include participants with Stage IIIC cutaneous melanoma, as defined by this classification scheme. Within each cohort, participants will be randomized (1:1 ratio) to receive vemurafenib or matching placebo over a 52-week period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma of cutaneous origin
* Participants with BRAFV600 mutation-positive, cutaneous melanoma (either pathologic Stage IIC or Stage III according to AJCC Staging Criteria version 7 that has been completely resected
* BRAF V600 mutation status of the current primary tumor or involved lymph node determined to be positive using the cobas BRAF V600 mutation test
* Surgically rendered free of disease within 90 days of randomization
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 5 years
* Fully recovered from the effects of any major surgery or significant traumatic injury prior to the first dose of study treatment
* Adequate hematologic, hepatic, and renal function

Exclusion Criteria:

* History of any systemic or local therapy (e.g., chemotherapy, biologic or targeted therapy, hormonal therapy, or photodynamic therapy) for the treatment or prevention of melanoma, including interferon alpha-2b and pegylated interferon alpha-2b
* History of limb perfusion therapy
* History of radiotherapy for the treatment of melanoma
* Invasive malignancy other than melanoma at the time of enrollment or within 5 years prior to first dose of study treatment
* Family history of inherited colon cancer syndromes
* Known personal history of >3 adenomatous colorectal polyps or a personal history of adenomatous colorectal polyp(s) >2 centimeters (cm) in size
* History of or current clinical, radiographic, or pathologic evidence of in-transit metastases, satellite, or microsatellite lesions
* History of or current clinical, radiographic, or pathologic evidence of recurrent lymph node involvement after resection of a primary melanoma with lymph node involvement at any time in the past
* History of local and/or regional and/or distant melanoma recurrence
* History or current radiographic or pathologic evidence of distant metastases
* History of clinically significant cardiac or pulmonary dysfunction
* Major surgical procedure or significant traumatic injury within 4 weeks prior to first dose of study treatment
* Infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2012-09-24 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2018-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (207):
- United States (47):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA Department of Medicine; Division of Hematology / Oncology, California City, California
  - Kaiser Permanente - Hayward, Hayward, California
  - UCLA Hematology Oncology - Irvine, Irvine, California
  - UCSD Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute - W LA Office, Los Angeles, California
  - Cancer Center Of Santa Barbara; Network Clinical Research Specialist, Los Angeles, California
  - TRIO-US Network Administration; Network Clinical Research Specialist, Los Angeles, California
  - Kaiser Foundation Hospital - Oakland (W. MacArthur), Oakland, California
  - Kaiser Permanente - Oakland, Oakland, California
  - UCLA Healthcare/Pasadena Oncology, Pasadena, California
  - Kaiser Permanente - Roseville, Roseville, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente, San Francisco, California
  - K. Permanente - San Jose, San Jose, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Kaiser Permanente - Santa Clara, Santa Clara, California
  - Kaiser Permanente - South San Francisco, South San Francisco, California
  - Stanford University School of Medicine; Stanford Hospital Pharmacy, Stanford, California
  - UCLA Cancer Center Hema/Oncol, Valencia, California
  - Kaiser Permanente - Vallejo, Vallejo, California
  - Kaiser Permanente - Walnut Creek, Walnut Creek, California
  - UCLA Hematology Oncology - Westlake, Westlake Village, California
  - University Of Colorado, Aurora, Colorado
  - St. Mary's Hospital Regional Cancer Center, Grand Junction, Colorado
  - Florida Cancer Specialists - Broadway, Fort Myers, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - GulfCoast Oncology, Sarasota, Florida
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Indiana University Health; Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University Department of Medicine; Division of Infectious Diseases, Indianapolis, Indiana
  - U of L - Physicians Pulmonology; Dept of Neuroradiology and Dept of Diagnostic Radiology, Louisville, Kentucky
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - St. Luke's Hospital, Kansas City, Missouri
  - University of Kansas Medical Center; Cancer Center, Kansas City, Missouri
  - Washington University; Dept of Medicine/Div of Medical Oncology, St Louis, Missouri
  - Atlantic Health Systems; Pediatrics, Randolph Township, New Jersey
  - New York University Medical Center PRIME; NYU Clinical Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center; Oncology, Durham, North Carolina
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - MUSC Hollings Cancer Center/cannon Park Place; Attn: Tamara Saunders, Charleston, South Carolina
  - West Clinic, Germantown, Tennessee
  - Tennessee Oncology PLLC - Nashville (20th Ave), Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Mary Babb Randolph Cancer Center, Morgantown, West Virginia
- Argentina (7):
  - Fundación CIDEA, Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Ciudad Autonoma Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Hospital Universitario Austral, Derqui-Pilar
  - Centro de Investigacion Pergamino SA, Pergamino
  - Instituto de Oncología de Rosario, Rosario
  - ISIS Clinica Especializada, Santa Fe
- Australia (15):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Border Medical Oncology, Wodonga, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Cairns Base Hospital, Cairns, Queensland
  - The Townsville Hospital; Townsville Cancer Centre, Townsville, Queensland
  - Royal Adelaide Hospital; Hepatology, Adelaide, South Australia
  - Queen Elizabeth Hospital, Woodville, South Australia
  - Launceston General Hospital; Gastroenterology Research, Launceston, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Peninsula Oncology Centre; Frankston Private, Frankston, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (4):
  - Medizinische Universität Innsbruck, Innsbruck
  - Krankenanstalt Rudolfstiftung Wien, Vienna
  - Medizinische Universität Wien, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (6):
  - ZNA Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - AZ Groeninge, Apotheek, Kortrijk
- Brazil (6):
  - Trymed Clinical Research, Belo Horizonte, Minas Gerais
  - CITO - Centro Integrado de Terapia Onco-Hematológica - Hospital da Cidade de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Clinica de Oncologia de Porto Alegre - CliniOnco, Porto Alegre, Rio Grande do Sul
  - Hospital de Caridade de Ijuí, Ijuí, Rondônia
  - Hospital Sírio-Libanês, São Paulo, São Paulo
- Canada (10):
  - BC Cancer Agency Vancouver Centre - PARENT; BC Cancer Agency, Vancouver, British Columbia
  - Saint Boniface General Hospital; Section of Nephrology BG 007, Winnipeg, Manitoba
  - Saint John Regional Hospital; Department of Oncology, Saint John, New Brunswick
  - LHSC - Victoria Hospital; Department of Pediatrics, London, Ontario
  - The Ottawa Hospital Cancer Center; General Campus, Ottawa, Ontario
  - Toronto Sunnybrook Hospital, Toronto, Ontario
  - Princess Margaret Hospital; Department of Med Oncology, Toronto, Ontario
  - CHUM Hôpital Notre-Dame, Montreal, Quebec
  - Mcgill University - Royal Victoria Hospital; Oncology, Montreal, Quebec
  - CHUQ - Hôtel-Dieu de Québec, Ste-Foy, Quebec
- Croatia (4):
  - General Hospital Pula, Pula
  - General Hospital Varazdin, Varaždin
  - Clinical Hospital Center Sestre Milosrdnice, Zagreb
  - Clinical Hospital Centre Zagreb, Zagreb
- Czechia (7):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultní nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Nemocnice Na Bulovce, Prague
- Estonia (3):
  - East Tallinn Central Hospital; Clinic of Internal Medicine, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital; Clinic of Hematology and Oncology, Tartu
- France (11):
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Groupe Hospitalier Saint André - Hôpital Saint André, Bordeaux
  - Hôpital Ambroise Paré - Boulogne-Billancourt; Respiratory, Boulogne-Billancourt
  - Hopital Claude Huriez - CHU Lille, Lille
  - Hopital de la Timone, Marseille
  - CHU NANTES - Hôtel Dieu; Pharmacy, Nantes
  - CHU Nice - Hopital de l'Archet 2, Nice
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Rouen Hopital; Service de Neurologie, Rouen
  - CHU de Toulouse - Hôpital Larrey, Toulouse
- Germany (12):
  - St. Josef-Hospital Universitaetsklinikum, Bochum
  - Elbekliniken Buxtehude GmbH, Buxtehude
  - Universitätsklinikum Koeln, Cologne
  - Universitätsklinikum Essen, Essen
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel; Klinik fuer Allgemeine Innere Medizin, Kiel
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz; Apotheke, Mainz
  - Klinikum Mannheim GmbH Universitätsklinikum, Mannheim
  - Fachklinik Hornheide, Münster
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Wurzburg, Würzburg
- Ireland (4):
  - Cork University Hospital, Cork
  - Mater Private Hospital, Dublin
  - The Mater Misericordiae Hospital, Dublin
  - University College Hospital, Galway
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (13):
  - Istituto Tumori Giovanni Paolo II IRCSS; Ospedale Oncologico Bari, Bari, Apulia
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome, Lazio
  - Istituto Nazionale Tumori Regina Elena IRCCS, Rome, Lazio
  - IDI-Istituto Dermopatico dell'Immacolata IRCCS, Rome, Lazio
  - Istituto Nazionale per la Ricerca sul Cancro di Genova, Genoa, Liguria
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo, Lombardy
  - Asst Degli Spedali Civili Di Brescia, Brescia, Lombardy
  - Ospedale San Raffaele, Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - IRCCS Istituto Clinico Humanitas; Farmacia, Rozzano, Lombardy
  - A.O.U. Senese Policlinico Santa Maria Alle Scotte, Siena, Tuscany
  - IOV - Istituto Oncologico Veneto IRCCS, Padua, Veneto
- Mexico (4):
  - Centro Oncologico Belenus, Cuernavaca
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - Centro Regiomontano de Investigación Clínica, Monterrey
  - Sanatorio la Luz, Morelia
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Leids Universitair Medisch Centrum; Cardiology, Leiden
- New Zealand (2):
  - Christchurch Hospital NZ, Christchurch
  - Wellington Hospital, Wellington
- Stavanger Universitetssykehus, Helse Stavanger HF, Stavanger, Norway
- Poland (4):
  - SPZOZ MSW zWarmińsko-MazurskimCen.Onko.wOlsztynie, Olsztyn
  - Przychodnia Med-Polonia Sp. z o.o., Poznan
  - Centrum Onkologii- Instytut; im. M.Skłodowskiej-Curie, Warsaw
  - Dolnoslaskie Centrum Onkologii, Wroclaw
- Portugal (4):
  - IPO de Coimbra; Servico de Oncologia Medica, Coimbra
  - Hospital do Espirito Santo; Servico de Oncologia Medica, Evora
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Russia (4):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Krasnodar City Oncology Center, Krasnodar
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow
  - Scientific Research Oncology Institute named after N.N. Petrov, Saint Petersburg
- Serbia (4):
  - Institute of Oncology and Radiology of Serbia, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Bezanijska Kosa, Belgrade
  - Institute for oncology of Vojvodina, Kamenitz
- South Africa (5):
  - GVI Rondebosch Oncology Centre, Cape Town
  - Mary Potter Oncology Centre, Groenkloof
  - Groote Schuur Hospital Radiation Oncology Department; Department of Radiation Oncology, Observatory
  - University of Pretoria Oncology Department, Pretoria
  - Sandton Oncology Medical Group, Sandton
- Spain (6):
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, LA Coruña
  - Hospital Costa del Sol; Servicio de Oncologia, Marbella, Malaga
  - Hospital de la Santa Creu; i Sant Pau, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (3):
  - Länssjukhuset Ryhov, Jönköping
  - Norrlands Universitetssjukhus, Umeå
  - Centrallasarettet Växjö, Vaxjo
- CHUV; Departement d'Oncologie, Lausanne, Switzerland
- Ukraine (2):
  - CI Dnipropetrovsk CMCH 4 of Dnipropetrovsk RC Dept of Chemotherapy SI Dnipropetrovsk MA of MOHU, Dnipropetrovsk
  - Lviv State Oncological Regional Treatment and Diagnostic Center, Lviv
- United Kingdom (10):
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - Queen Elizabeth Hospital, Kings Lynn
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - Nottingham University Hospitals City Campus, Nottingham
  - Churchill Hospital, Oxford
  - Royal Cornwall Hospital, Truro
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Ascierto PA, Lewis KD, Di Giacomo AM, Demidov L, Mandala M, Bondarenko I, Herbert C, Mackiewicz A, Rutkowski P, Guminski A, Simmons B, Ye C, Hooper G, Wongchenko MJ, Goodman GR, Yan Y, Schadendorf D. Prognostic impact of baseline tumour immune infiltrate on disease-free survival in patients with completely resected, BRAFv600 mutation-positive melanoma receiving adjuvant vemurafenib. Ann Oncol. 2020 Jan;31(1):153-159. doi: 10.1016/j.annonc.2019.10.002. PMID 31912791
- [Derived] Maio M, Lewis K, Demidov L, Mandala M, Bondarenko I, Ascierto PA, Herbert C, Mackiewicz A, Rutkowski P, Guminski A, Goodman GR, Simmons B, Ye C, Yan Y, Schadendorf D; BRIM8 Investigators. Adjuvant vemurafenib in resected, BRAFV600 mutation-positive melanoma (BRIM8): a randomised, double-blind, placebo-controlled, multicentre, phase 3 trial. Lancet Oncol. 2018 Apr;19(4):510-520. doi: 10.1016/S1470-2045(18)30106-2. Epub 2018 Feb 21. PMID 29477665

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 Vemurafenib | Cohort 1 Placebo | Cohort 2 Vemurafenib | Cohort 2 Placebo
Started | 157 | 157 | 93 | 91
Completed | 114 | 110 | 57 | 52
Not Completed | 43 | 47 | 36 | 39
Not completed — Reason Not Specified | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 8 | 9 | 8
Not completed — Non-compliance | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 7 | 6 | 2 | 4
Not completed — Death | 18 | 33 | 25 | 26

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants enrolled in the study, whether or not they had received study medication.
Groups:
- Cohort 1 Vemurafenib: Participants with completely resected Stage IIC, IIIA, or IIIB cutaneous melanoma) received vemurafenib, 960 mg twice daily, in 28-day cycles, for up to 52 weeks
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Vemurafenib | Cohort 1 Placebo | Cohort 2 Vemurafenib | Cohort 2 Placebo | Total
Number analyzed (Participants) | 157 | 157 | 93 | 91 | 498
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The intent-to-treat (ITT) population included all participants enrolled in the study, whether or not they had received study medication.
  years | 50.7 (12.4) | 49.6 (12.7) | 51.6 (14.1) | 49.1 (12.9) | 50.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The intent-to-treat (ITT) population included all participants enrolled in the study, whether or not they had received study medication.
  Participants
    Female | 73 | 69 | 41 | 32 | 215
    Male | 84 | 88 | 52 | 59 | 283
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The intent-to-treat (ITT) population included all participants enrolled in the study, whether or not they had received study medication.
  Participants
    Hispanic or Latino | 12 | 2 | 8 | 3 | 25
    Not Hispanic or Latino | 138 | 148 | 79 | 80 | 445
    Unknown or Not Reported | 7 | 7 | 6 | 8 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The intent-to-treat (ITT) population included all participants enrolled in the study, whether or not they had received study medication.
  Participants
    White | 150 | 150 | 84 | 81 | 465
    Other | 1 | 2 | 1 | 2 | 6
    Multiple | 0 | 0 | 1 | 0 | 1
    Unknown | 6 | 5 | 7 | 8 | 26

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival (DFS) as Assessed Using Contrast-Enhanced Magnetic Resonance Imaging (MRI) or Contrast Enhanced Computed Tomography (CT)
Description: DFS was defined as the time from randomization until the date of the first local, regional, or distant melanoma recurrence, occurrence of new primary melanoma, or death from any cause.
Time Frame: From randomization until the date of the first local, regional, or distant melanoma recurrence, occurrence of new primary melanoma, or death from any cause (up to the April 17, 2017 data cut-off, approximately 4.5 years)
Population: The ITT population included all participants enrolled in the study, whether or not they had received study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 Vemurafenib | Cohort 1 Placebo | Cohort 2 Vemurafenib | Cohort 2 Placebo
Number analyzed (Participants) | 157 | 157 | 93 | 91
months | NA [NA to NA] — Not estimable due to low number of events. | 36.9 [21.4 to NA] — Not estimable due to low number of events. | 23.1 [18.6 to 26.5] | 15.4 [11.1 to 35.9]
Statistical Analysis 1: Comparison: Cohort 1 Vemurafenib vs Cohort 1 Placebo; Test type: Superiority; p = 0.0010, Log Rank; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.37 to 0.78]
Statistical Analysis 2: Comparison: Cohort 2 Vemurafenib vs Cohort 2 Placebo; Test type: Superiority; p = 0.2598, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.54 to 1.18]

2. Secondary Outcome: Distant Metastasis-Free Survival (DMFS) as Assessed Using Contrast-Enhanced MRI or Contrast Enhanced CT
Description: DMFS was defined as the time from randomization until the date of diagnosis of distant (i.e. non-locoregional) metastases or death from any cause.
Time Frame: From randomization until the date of diagnosis of distant (i.e., non-locoregional) metastases or death from any cause (up to the April 17, 2017 data cut-off, approximately 4.5 years)
Population: The ITT population included all participants enrolled in the study, whether or not they had received study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 Vemurafenib | Cohort 1 Placebo | Cohort 2 Vemurafenib | Cohort 2 Placebo
Number analyzed (Participants) | 157 | 157 | 93 | 91
months | NA [NA to NA] — Not estimable due to low number of events. | NA [36.9 to NA] — Not estimable due to low number of events. | 37.2 [22.1 to NA] — Not estimable due to low number of events. | 30.7 [24.5 to NA] — Not estimable due to low number of events.
Statistical Analysis 1: Comparison: Cohort 1 Vemurafenib vs Cohort 1 Placebo; Test type: Superiority; p = 0.0133, Log Rank; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.37 to 0.90]
Statistical Analysis 2: Comparison: Cohort 2 Vemurafenib vs Cohort 2 Placebo; Test type: Superiority; p = 0.6815, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.57 to 1.44]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization until the date of death from any cause.
Time Frame: From randomization until the date of death from any cause (up until 13-July-2018, approximately 6 years)
Population: The ITT population included all participants enrolled in the study, whether or not they had received study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 Vemurafenib | Cohort 1 Placebo | Cohort 2 Vemurafenib | Cohort 2 Placebo
Number analyzed (Participants) | 157 | 157 | 93 | 91
months | NA [60 to NA] — Not estimable due to low number of events. | NA [NA to NA] — Not estimable due to low number of events. | 59.9 [54.6 to 59.9] | NA [52.6 to NA] — Not estimable due to low number of events.
Statistical Analysis 1: Comparison: Cohort 1 Vemurafenib vs Cohort 1 Placebo; Test type: Superiority; p = 0.0274, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.30 to .94]
Statistical Analysis 2: Comparison: Cohort 2 Vemurafenib vs Cohort 2 Placebo; Test type: Superiority; p = 0.8597, Log Rank; Hazard Ratio (HR) = .95, 95% CI 2-sided [0.55 to 1.66]

4. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution.
Time Frame: From randomization up to study completion or discontinuation (up until 13-July-2018, approximately 6 years)
Population: The safety population included all participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 Vemurafenib | Cohort 1 Placebo | Cohort 2 Vemurafenib | Cohort 2 Placebo
Number analyzed (Participants) | 154 | 156 | 93 | 91
percentage of participants | 99.4 | 88.5 | 100.0 | 89.0

5. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) 30-Item Quality of Life Questionnaire (QLQ-C30) Score
Description: European Organisation for Research and Treatment of Cancer 30-Item Quality of Life Questionnaire assesses 8 symptoms, function, financial difficulties, and a global health status/health-related quality of life (HRQoL). Most questions use a 4-point scale (1 'Not at all' to 4 'Very much';2 questions use a 7-point scale (1 'very poor' to 7 'Excellent'). Scores were averaged and transformed to a 0-100 scale. Higher scores for the function and HRQoL represent higher levels of functioning and HRQoL, higher scores for the symptom represent higher levels of symptoms/problems, higher score for financial difficulty represent higher level of perceived financial burden of treatment. Changes of 5-10 points are considered to represent a minimally important difference to participants. A positive value means an increase, and negative value means a decrease in score at the indicated time-point relative to the score at baseline (Cycle 1 Day 1).
Time Frame: Day 1, Day 8, Day 15, Day 22 of Cycle 1;Day 1, Day 15 of Cycle 2;Day 1 Cycles 3-13;end of treatment(up to 13 months);every 13 weeks thereafter until recurrence or occurrence of a new primary melanoma (up to 17-Apr-17 data cut-off,approximately 4.5 years)
Population: The patient-reported outcome (PRO)-evaluable population included all participants who received at least one dose of vemurafenib and who had both a baseline assessment and at least one post-baseline QLQ-C30 assessment that generated a score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 Vemurafenib | Cohort 1 Placebo | Cohort 2 Vemurafenib | Cohort 2 Placebo
Number analyzed (Participants) | 138 | 147 | 87 | 89
score on a scale
  Appetite Loss: Cycle 1 Day 1 (Baseline): number analyzed (Participants) | 138 | 147 | 86 | 89
  Appetite Loss: Cycle 1 Day 1 (Baseline) | 3.6 (11.2) | 3.9 (14.9) | 3.5 (10.3) | 3.4 (11.3)
  Appetite Loss: Change at Cycle 1 Day 8: number analyzed (Participants) | 24 | 22 | 16 | 19
  Appetite Loss: Change at Cycle 1 Day 8 | 2.8 (9.4) | 1.5 (7.1) | 10.4 (16.0) | 0.0 (11.1)
  Appetite Loss: Change at Cycle 1 Day 15: number analyzed (Participants) | 132 | 139 | 79 | 84
  Appetite Loss: Change at Cycle 1 Day 15 | 16.7 (26.5) | 1.4 (12.0) | 12.2 (22.8) | 1.2 (17.5)
  Appetite Loss: Change at Cycle 1 Day 22: number analyzed (Participants) | 22 | 21 | 15 | 17
  Appetite Loss: Change at Cycle 1 Day 22 | 7.6 (14.3) | 3.2 (10.0) | 11.1 (20.6) | 3.9 (20.0)
  Appetite Loss: Change at Cycle 2 Day 1: number analyzed (Participants) | 126 | 142 | 82 | 84
  Appetite Loss: Change at Cycle 2 Day 1 | 9.5 (21.0) | 1.2 (10.1) | 12.2 (23.7) | 1.6 (15.4)
  Appetite Loss: Change at Cycle 2 Day 15: number analyzed (Participants) | 119 | 134 | 79 | 81
  Appetite Loss: Change at Cycle 2 Day 15 | 9.5 (22.2) | 1.0 (12.2) | 6.8 (16.3) | 0.8 (14.9)
  Appetite Loss: Change at Cycle 3 Day 1: number analyzed (Participants) | 119 | 129 | 80 | 77
  Appetite Loss: Change at Cycle 3 Day 1 | 10.4 (20.7) | 1.6 (10.1) | 8.3 (18.0) | 0.4 (14.8)
  Appetite Loss: Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 129 | 78 | 76
  Appetite Loss: Change at Cycle 4 Day 1 | 9.5 (20.9) | 1.3 (12.1) | 10.3 (20.3) | 2.6 (15.2)
  Appetite Loss: Change at Cycle 5 Day 1: number analyzed (Participants) | 110 | 117 | 72 | 64
  Appetite Loss: Change at Cycle 5 Day 1 | 13.3 (23.5) | 1.4 (12.7) | 7.4 (15.0) | -0.5 (12.6)
  Appetite Loss: Change at Cycle 6 Day 1: number analyzed (Participants) | 106 | 112 | 69 | 63
  Appetite Loss: Change at Cycle 6 Day 1 | 9.7 (21.1) | 2.4 (12.4) | 13.0 (21.6) | 1.1 (17.9)
  Appetite Loss: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 108 | 68 | 59
  Appetite Loss: Change at Cycle 7 Day 1 | 10.7 (22.8) | 1.5 (14.0) | 7.4 (16.1) | 4.0 (18.7)
  Appetite Loss: Change at Cycle 8 Day 1: number analyzed (Participants) | 105 | 105 | 65 | 53
  Appetite Loss: Change at Cycle 8 Day 1 | 10.2 (22.7) | 1.9 (13.7) | 10.8 (18.7) | -0.6 (12.2)
  Appetite Loss: Change at Cycle 9 Day 1: number analyzed (Participants) | 100 | 101 | 63 | 52
  Appetite Loss: Change at Cycle 9 Day 1 | 9.7 (25.2) | 2.3 (13.5) | 7.9 (17.7) | 3.8 (15.7)
  Appetite Loss: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 63 | 47
  Appetite Loss: Change at Cycle 10 Day 1 | 7.3 (18.9) | 1.7 (15.5) | 4.8 (15.7) | 0.0 (12.0)
  Appetite Loss: Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 93 | 57 | 48
  Appetite Loss: Change at Cycle 11 Day 1 | 5.4 (19.2) | 1.8 (14.2) | 4.7 (13.3) | 0.7 (12.8)
  Appetite Loss: Change at Cycle 12 Day 1: number analyzed (Participants) | 90 | 91 | 55 | 48
  Appetite Loss: Change at Cycle 12 Day 1 | 8.5 (20.9) | 1.5 (14.0) | 7.3 (15.3) | 0.0 (11.9)
  Appetite Loss: Change at Cycle 13 Day 1: number analyzed (Participants) | 82 | 89 | 54 | 45
  Appetite Loss: Change at Cycle 13 Day 1 | 5.7 (17.2) | 1.9 (13.6) | 6.2 (14.6) | 0.7 (11.2)
  Appetite Loss: Change at End of Treatment: number analyzed (Participants) | 123 | 125 | 66 | 75
  Appetite Loss: Change at End of Treatment | 2.7 (16.3) | 0.8 (20.1) | 5.1 (18.7) | 2.7 (18.8)
  Appetite Loss: Change at PT 13 Weeks: number analyzed (Participants) | 90 | 74 | 55 | 38
  Appetite Loss: Change at PT 13 Weeks | 0.0 (13.2) | 1.8 (16.5) | -1.2 (6.3) | 1.8 (10.8)
  Appetite Loss: Change at PT 26 Weeks: number analyzed (Participants) | 90 | 72 | 47 | 35
  Appetite Loss: Change at PT 26 Weeks | 0.7 (16.6) | -1.4 (15.3) | 3.5 (17.4) | 1.0 (12.7)
  Appetite Loss: Change at PT 39 Weeks: number analyzed (Participants) | 79 | 68 | 42 | 33
  Appetite Loss: Change at PT 39 Weeks | -0.4 (12.5) | -0.5 (7.0) | -0.8 (9.0) | 2.0 (14.3)
  Appetite Loss: Change at PT 52 Weeks: number analyzed (Participants) | 76 | 62 | 26 | 25
  Appetite Loss: Change at PT 52 Weeks | 0.4 (17.6) | 0.0 (12.1) | -1.3 (6.5) | 2.7 (9.2)
  Appetite Loss: Change at PT 65 Weeks: number analyzed (Participants) | 53 | 38 | 17 | 18
  Appetite Loss: Change at PT 65 Weeks | -1.9 (12.1) | 0.9 (14.5) | 0.0 (0.0) | 5.6 (17.1)
  Appetite Loss: Change at PT 78 Weeks: number analyzed (Participants) | 46 | 33 | 15 | 9
  Appetite Loss: Change at PT 78 Weeks | -0.7 (11.1) | 2.0 (14.3) | 0.0 (0.0) | 3.7 (11.1)
  Appetite Loss: Change at PT 91 Weeks: number analyzed (Participants) | 32 | 29 | 15 | 12
  Appetite Loss: Change at PT 91 Weeks | 2.1 (16.8) | 2.3 (12.4) | 0.0 (0.0) | 2.8 (9.6)
  Appetite Loss: Change at PT 104 Weeks: number analyzed (Participants) | 27 | 25 | 10 | 9
  Appetite Loss: Change at PT 104 Weeks | -1.2 (11.3) | -1.3 (6.7) | 0.0 (0.0) | -3.7 (11.1)
  Appetite Loss: Change at PT 117 Weeks: number analyzed (Participants) | 22 | 17 | 9 | 5
  Appetite Loss: Change at PT 117 Weeks | -1.5 (12.5) | 2.0 (14.3) | 0.0 (0.0) | 0.0 (0.0)
  Appetite Loss: Change at PT 130 Weeks: number analyzed (Participants) | 17 | 12 | 5 | 5
  Appetite Loss: Change at PT 130 Weeks | 0.0 (0.0) | 2.8 (17.2) | 0.0 (0.0) | 0.0 (0.0)
  Appetite Loss: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Appetite Loss: Change at PT 143 Weeks | -4.8 (12.6) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Appetite Loss: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Appetite Loss: Change at PT 156 Weeks | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  | 16.7 (23.6)
  Appetite Loss: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Appetite Loss: Change at PT 169 Weeks | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Appetite Loss: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Appetite Loss: Change at PT 182 Weeks | 0.0 (0.0) |  |  |
  Appetite Loss: Change at PT/Discontinuation: number analyzed (Participants) | 8 | 1 | 6 | 1
  Appetite Loss: Change at PT/Discontinuation | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable.
  Cognitive Functioning: Cycle 1 Day 1 (Baseline) | 93.0 (14.1) | 92.0 (16.2) | 91.4 (17.2) | 94.9 (11.6)
  Cognitive Functioning: Change at Cycle 1 Day 8: number analyzed (Participants) | 24 | 22 | 16 | 19
  Cognitive Functioning: Change at Cycle 1 Day 8 | -2.1 (12.3) | 1.5 (14.5) | 0.0 (10.5) | 2.6 (6.2)
  Cognitive Functioning: Change at Cycle 1 Day 15: number analyzed (Participants) | 132 | 139 | 78 | 84
  Cognitive Functioning: Change at Cycle 1 Day 15 | -4.3 (13.1) | 0.8 (12.6) | -3.8 (13.4) | -0.8 (11.5)
  Cognitive Functioning: Change at Cycle 1 Day 22: number analyzed (Participants) | 22 | 21 | 15 | 17
  Cognitive Functioning: Change at Cycle 1 Day 22 | -0.8 (17.4) | 1.6 (11.7) | -3.3 (9.3) | -4.9 (14.1)
  Cognitive Functioning: Change at Cycle 2 Day 1: number analyzed (Participants) | 127 | 142 | 82 | 84
  Cognitive Functioning: Change at Cycle 2 Day 1 | -2.4 (14.2) | -2.5 (14.3) | -2.2 (12.2) | 0.0 (13.9)
  Cognitive Functioning: Change at Cycle 2 Day 15: number analyzed (Participants) | 119 | 134 | 80 | 80
  Cognitive Functioning: Change at Cycle 2 Day 15 | -3.8 (15.1) | -1.1 (14.6) | -3.1 (11.9) | -0.4 (15.2)
  Cognitive Functioning: Change at Cycle 3 Day 1: number analyzed (Participants) | 119 | 129 | 81 | 78
  Cognitive Functioning: Change at Cycle 3 Day 1 | -3.6 (13.4) | -0.6 (12.0) | -2.5 (12.4) | -2.1 (13.3)
  Cognitive Functioning: Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 129 | 78 | 76
  Cognitive Functioning: Change at Cycle 4 Day 1 | -3.8 (14.6) | -1.3 (15.1) | -4.9 (13.5) | -2.9 (13.7)
  Cognitive Functioning: Change at Cycle 5 Day 1: number analyzed (Participants) | 110 | 116 | 72 | 64
  Cognitive Functioning: Change at Cycle 5 Day 1 | -6.2 (17.3) | -2.0 (14.9) | -3.9 (12.7) | -3.6 (15.3)
  Cognitive Functioning: Change at Cycle 6 Day 1: number analyzed (Participants) | 106 | 112 | 69 | 63
  Cognitive Functioning: Change at Cycle 6 Day 1 | -5.7 (15.8) | -2.1 (12.5) | -4.1 (16.0) | -3.4 (18.2)
  Cognitive Functioning: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 108 | 68 | 59
  Cognitive Functioning: Change at Cycle 7 Day 1 | -6.3 (17.3) | -3.1 (13.3) | -3.9 (15.5) | -5.6 (15.0)
  Cognitive Functioning: Change at Cycle 8 Day 1: number analyzed (Participants) | 104 | 106 | 65 | 53
  Cognitive Functioning: Change at Cycle 8 Day 1 | -7.4 (16.1) | -3.6 (16.9) | -5.1 (16.6) | -4.7 (13.2)
  Cognitive Functioning: Change at Cycle 9 Day 1: number analyzed (Participants) | 100 | 101 | 63 | 52
  Cognitive Functioning: Change at Cycle 9 Day 1 | -8.2 (18.1) | -4.6 (17.3) | -5.8 (17.7) | -5.4 (12.2)
  Cognitive Functioning: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 63 | 47
  Cognitive Functioning: Change at Cycle 10 Day 1 | -9.0 (20.1) | -3.6 (17.4) | -4.5 (17.5) | -8.2 (19.3)
  Cognitive Functioning: Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 93 | 57 | 48
  Cognitive Functioning: Change at Cycle 11 Day 1 | -10.6 (20.1) | -2.9 (15.9) | -5.0 (15.1) | -3.8 (12.5)
  Cognitive Functioning: Change at Cycle 12 Day 1: number analyzed (Participants) | 90 | 91 | 55 | 48
  Cognitive Functioning: Change at Cycle 12 Day 1 | -8.7 (21.5) | -4.0 (14.6) | -3.9 (13.6) | -4.5 (14.5)
  Cognitive Functioning: Change at Cycle 13 Day 1: number analyzed (Participants) | 82 | 89 | 54 | 45
  Cognitive Functioning: Change at Cycle 13 Day 1 | -7.7 (20.7) | -3.9 (16.1) | -6.5 (15.7) | -5.2 (12.7)
  Cognitive Functioning: Change at End of Treatment: number analyzed (Participants) | 123 | 125 | 67 | 75
  Cognitive Functioning: Change at End of Treatment | -4.9 (17.3) | -3.5 (19.5) | -4.0 (17.2) | -6.9 (14.3)
  Cognitive Functioning: Change at PT 13 Weeks: number analyzed (Participants) | 90 | 74 | 56 | 38
  Cognitive Functioning: Change at PT 13 Weeks | -4.4 (14.9) | -1.6 (14.1) | -1.5 (14.0) | -3.5 (14.1)
  Cognitive Functioning: Change at PT 26 Weeks: number analyzed (Participants) | 90 | 72 | 47 | 35
  Cognitive Functioning: Change at PT 26 Weeks | -2.8 (16.2) | -2.5 (14.2) | -2.1 (15.4) | -3.8 (13.5)
  Cognitive Functioning: Change at PT 39 Weeks: number analyzed (Participants) | 79 | 68 | 41 | 33
  Cognitive Functioning: Change at PT 39 Weeks | -2.1 (13.2) | -1.0 (14.6) | -2.0 (11.9) | -3.0 (11.4)
  Cognitive Functioning: Change at PT 52 Weeks: number analyzed (Participants) | 76 | 62 | 27 | 25
  Cognitive Functioning: Change at PT 52 Weeks | -3.5 (17.3) | -1.9 (9.1) | 1.2 (13.0) | -7.3 (12.8)
  Cognitive Functioning: Change at PT 65 Weeks: number analyzed (Participants) | 53 | 38 | 17 | 18
  Cognitive Functioning: Change at PT 65 Weeks | -4.4 (17.3) | -3.9 (15.2) | -1.0 (12.5) | -4.6 (11.2)
  Cognitive Functioning: Change at PT 78 Weeks: number analyzed (Participants) | 46 | 33 | 15 | 9
  Cognitive Functioning: Change at PT 78 Weeks | -2.5 (17.2) | -3.5 (19.4) | -1.1 (14.7) | -7.4 (12.1)
  Cognitive Functioning: Change at PT 91 Weeks: number analyzed (Participants) | 33 | 29 | 15 | 12
  Cognitive Functioning: Change at PT 91 Weeks | -2.5 (16.2) | -2.3 (15.9) | 3.3 (11.3) | -5.6 (13.0)
  Cognitive Functioning: Change at PT 104 Weeks: number analyzed (Participants) | 27 | 25 | 10 | 9
  Cognitive Functioning: Change at PT 104 Weeks | 1.2 (14.6) | -4.0 (16.9) | 3.3 (13.1) | -5.6 (11.8)
  Cognitive Functioning: Change at PT 117 Weeks: number analyzed (Participants) | 22 | 17 | 8 | 5
  Cognitive Functioning: Change at PT 117 Weeks | 1.5 (12.5) | 0.0 (10.2) | -2.1 (5.9) | -6.7 (14.9)
  Cognitive Functioning: Change at PT 130 Weeks: number analyzed (Participants) | 17 | 12 | 5 | 5
  Cognitive Functioning: Change at PT 130 Weeks | -3.9 (15.1) | -1.4 (15.0) | 0.0 (0.0) | -6.7 (14.9)
  Cognitive Functioning: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Cognitive Functioning: Change at PT 143 Weeks | 4.8 (18.5) | 0.0 (0.0) | 0.0 (0.0) | -8.3 (11.8)
  Cognitive Functioning: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Cognitive Functioning: Change at PT 156 Weeks | 11.1 (19.2) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  | -16.7 (23.6)
  Cognitive Functioning: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Cognitive Functioning: Change at PT 169 Weeks | 16.7 (23.6) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Cognitive Functioning: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Cognitive Functioning: Change at PT 182 Weeks | 11.1 (19.2) |  |  |
  Cognitive Functioning: Change at PT/Discontin.: number analyzed (Participants) | 8 | 1 | 6 | 1
  Cognitive Functioning: Change at PT/Discontin. | -2.1 (16.5) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. | -5.6 (8.6) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable.
  Constipation: Cycle 1 Day 1 (Baseline): number analyzed (Participants) | 138 | 146 | 87 | 88
  Constipation: Cycle 1 Day 1 (Baseline) | 3.1 (10.6) | 5.7 (16.3) | 4.6 (12.6) | 5.7 (15.3)
  Constipation: Change at Cycle 1 Day 8: number analyzed (Participants) | 23 | 22 | 16 | 19
  Constipation: Change at Cycle 1 Day 8 | -2.9 (13.9) | 0.0 (0.0) | -2.1 (8.3) | -5.3 (12.5)
  Constipation: Change at Cycle 1 Day 15: number analyzed (Participants) | 130 | 138 | 80 | 83
  Constipation: Change at Cycle 1 Day 15 | 2.1 (17.0) | 0.7 (13.0) | 1.7 (13.9) | -0.4 (16.9)
  Constipation: Change at Cycle 1 Day 22: number analyzed (Participants) | 21 | 21 | 15 | 17
  Constipation: Change at Cycle 1 Day 22 | -1.6 (19.7) | 1.6 (7.3) | 0.0 (12.6) | -3.9 (16.2)
  Constipation: Change at Cycle 2 Day 1: number analyzed (Participants) | 124 | 141 | 82 | 83
  Constipation: Change at Cycle 2 Day 1 | 1.1 (12.7) | 1.4 (10.4) | 1.6 (13.8) | -0.4 (16.9)
  Constipation: Change at Cycle 2 Day 15: number analyzed (Participants) | 117 | 133 | 79 | 79
  Constipation: Change at Cycle 2 Day 15 | 1.4 (14.8) | 0.0 (13.0) | 0.0 (11.9) | -1.3 (15.5)
  Constipation: Change at Cycle 3 Day 1: number analyzed (Participants) | 115 | 127 | 79 | 77
  Constipation: Change at Cycle 3 Day 1 | -1.2 (12.4) | 1.0 (13.9) | 0.4 (12.5) | -1.7 (18.7)
  Constipation: Change at Cycle 4 Day 1: number analyzed (Participants) | 118 | 127 | 78 | 75
  Constipation: Change at Cycle 4 Day 1 | 0.6 (11.5) | 0.5 (16.8) | 0.0 (10.7) | -2.2 (14.8)
  Constipation: Change at Cycle 5 Day 1: number analyzed (Participants) | 107 | 116 | 71 | 64
  Constipation: Change at Cycle 5 Day 1 | -0.6 (9.1) | 0.3 (16.7) | 3.8 (14.4) | -3.1 (17.5)
  Constipation: Change at Cycle 6 Day 1: number analyzed (Participants) | 104 | 112 | 68 | 63
  Constipation: Change at Cycle 6 Day 1 | 0.6 (13.1) | 1.8 (16.6) | 5.4 (16.9) | -3.7 (20.0)
  Constipation: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 108 | 67 | 59
  Constipation: Change at Cycle 7 Day 1 | 3.1 (18.1) | 1.5 (19.0) | 3.0 (12.6) | -4.0 (15.3)
  Constipation: Change at Cycle 8 Day 1: number analyzed (Participants) | 103 | 106 | 64 | 53
  Constipation: Change at Cycle 8 Day 1 | 1.9 (14.6) | 1.6 (16.2) | 4.2 (15.1) | -1.9 (17.8)
  Constipation: Change at Cycle 9 Day 1: number analyzed (Participants) | 97 | 101 | 62 | 52
  Constipation: Change at Cycle 9 Day 1 | 1.4 (11.7) | -2.3 (13.5) | 3.2 (14.4) | -0.6 (20.3)
  Constipation: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 62 | 47
  Constipation: Change at Cycle 10 Day 1 | 1.4 (10.7) | -1.4 (12.7) | 1.6 (11.2) | -4.3 (17.9)
  Constipation: Change at Cycle 11 Day 1: number analyzed (Participants) | 92 | 93 | 56 | 48
  Constipation: Change at Cycle 11 Day 1 | 2.2 (14.7) | 0.0 (16.3) | 2.4 (14.0) | -4.9 (15.4)
  Constipation: Change at Cycle 12 Day 1: number analyzed (Participants) | 90 | 91 | 54 | 48
  Constipation: Change at Cycle 12 Day 1 | 4.8 (19.1) | -1.8 (14.4) | 3.1 (13.4) | -3.5 (14.2)
  Constipation: Change at Cycle 13 Day 1: number analyzed (Participants) | 81 | 89 | 54 | 45
  Constipation: Change at Cycle 13 Day 1 | 4.1 (18.5) | 0.0 (18.8) | 0.0 (11.2) | -3.7 (19.1)
  Constipation: Change at End of Treatment: number analyzed (Participants) | 122 | 124 | 67 | 74
  Constipation: Change at End of Treatment | 3.3 (15.1) | 2.4 (19.1) | 4.5 (17.3) | -1.4 (17.8)
  Constipation: Change at PT 13 Weeks: number analyzed (Participants) | 88 | 74 | 56 | 38
  Constipation: Change at PT 13 Weeks | 0.4 (17.1) | -0.5 (17.0) | 6.0 (16.9) | 0.9 (21.2)
  Constipation: Change at PT 26 Weeks: number analyzed (Participants) | 89 | 71 | 47 | 35
  Constipation: Change at PT 26 Weeks | -0.4 (13.8) | -0.9 (13.8) | 2.8 (9.4) | -1.0 (18.9)
  Constipation: Change at PT 39 Weeks: number analyzed (Participants) | 77 | 67 | 41 | 33
  Constipation: Change at PT 39 Weeks | 0.4 (14.8) | -0.5 (13.6) | 2.4 (13.7) | -4.0 (16.2)
  Constipation: Change at PT 52 Weeks: number analyzed (Participants) | 75 | 62 | 27 | 25
  Constipation: Change at PT 52 Weeks | 0.0 (13.4) | 0.0 (14.8) | 0.0 (9.2) | 0.0 (13.6)
  Constipation: Change at PT 65 Weeks: number analyzed (Participants) | 53 | 37 | 17 | 18
  Constipation: Change at PT 65 Weeks | 3.8 (14.1) | 3.6 (21.9) | 2.0 (14.3) | 0.0 (11.4)
  Constipation: Change at PT 78 Weeks: number analyzed (Participants) | 46 | 33 | 15 | 9
  Constipation: Change at PT 78 Weeks | -1.4 (9.8) | 6.1 (25.6) | 0.0 (0.0) | 0.0 (0.0)
  Constipation: Change at PT 91 Weeks: number analyzed (Participants) | 31 | 28 | 15 | 12
  Constipation: Change at PT 91 Weeks | -4.3 (11.4) | 6.0 (18.3) | 2.2 (8.6) | 0.0 (14.2)
  Constipation: Change at PT 104 Weeks: number analyzed (Participants) | 26 | 25 | 10 | 9
  Constipation: Change at PT 104 Weeks | 1.3 (14.8) | 4.0 (14.7) | -3.3 (10.5) | 0.0 (16.7)
  Constipation: Change at PT 117 Weeks: number analyzed (Participants) | 20 | 17 | 9 | 5
  Constipation: Change at PT 117 Weeks | -6.7 (13.7) | 9.8 (19.6) | 0.0 (0.0) | -6.7 (14.9)
  Constipation: Change at PT 130 Weeks: number analyzed (Participants) | 16 | 12 | 5 | 5
  Constipation: Change at PT 130 Weeks | -8.3 (14.9) | 5.6 (13.0) | 0.0 (23.6) | -6.7 (14.9)
  Constipation: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Constipation: Change at PT 143 Weeks | -9.5 (16.3) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Constipation: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Constipation: Change at PT 156 Weeks | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  | -16.7 (23.6)
  Constipation: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Constipation: Change at PT 169 Weeks | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Constipation: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Constipation: Change at PT 182 Weeks | -11.1 (19.2) |  |  |
  Constipation: Change at PT/Discontinuation: number analyzed (Participants) | 8 | 1 | 6 | 1
  Constipation: Change at PT/Discontinuation | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable.
  Diarrhoea: Cycle 1 Day 1 (Baseline) | 4.1 (13.0) | 5.4 (17.5) | 3.8 (13.9) | 4.1 (16.5)
  Diarrhoea: Change at Cycle 1 Day 8: number analyzed (Participants) | 24 | 22 | 16 | 19
  Diarrhoea: Change at Cycle 1 Day 8 | 4.2 (11.3) | 0.0 (10.3) | -4.2 (20.6) | -8.8 (24.4)
  Diarrhoea: Change at Cycle 1 Day 15: number analyzed (Participants) | 132 | 139 | 77 | 84
  Diarrhoea: Change at Cycle 1 Day 15 | 2.5 (21.3) | -0.7 (14.7) | 1.7 (19.4) | -1.6 (17.1)
  Diarrhoea: Change at Cycle 1 Day 22: number analyzed (Participants) | 22 | 21 | 15 | 17
  Diarrhoea: Change at Cycle 1 Day 22 | 3.0 (9.8) | -1.6 (16.6) | -2.2 (23.5) | -9.8 (25.7)
  Diarrhoea: Change at Cycle 2 Day 1: number analyzed (Participants) | 127 | 142 | 82 | 84
  Diarrhoea: Change at Cycle 2 Day 1 | 1.3 (19.9) | -0.9 (16.3) | 4.9 (21.7) | 0.0 (20.0)
  Diarrhoea: Change at Cycle 2 Day 15: number analyzed (Participants) | 119 | 134 | 80 | 80
  Diarrhoea: Change at Cycle 2 Day 15 | 1.7 (21.2) | -1.5 (19.1) | 0.4 (17.2) | 0.0 (16.8)
  Diarrhoea: Change at Cycle 3 Day 1: number analyzed (Participants) | 119 | 129 | 81 | 78
  Diarrhoea: Change at Cycle 3 Day 1 | 3.4 (21.9) | -0.3 (18.4) | 3.3 (19.4) | -0.9 (15.2)
  Diarrhoea: Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 129 | 78 | 76
  Diarrhoea: Change at Cycle 4 Day 1 | 3.9 (23.0) | 0.3 (19.8) | 5.6 (18.2) | -2.6 (18.7)
  Diarrhoea: Change at Cycle 5 Day 1: number analyzed (Participants) | 110 | 116 | 72 | 64
  Diarrhoea: Change at Cycle 5 Day 1 | 7.6 (23.7) | -1.4 (20.3) | 2.8 (20.0) | -3.6 (18.9)
  Diarrhoea: Change at Cycle 6 Day 1: number analyzed (Participants) | 106 | 112 | 69 | 63
  Diarrhoea: Change at Cycle 6 Day 1 | 7.2 (25.2) | -0.6 (20.0) | 7.2 (24.8) | -2.6 (19.2)
  Diarrhoea: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 108 | 68 | 59
  Diarrhoea: Change at Cycle 7 Day 1 | 9.4 (24.2) | -1.5 (21.6) | 4.9 (22.5) | -4.5 (18.0)
  Diarrhoea: Change at Cycle 8 Day 1: number analyzed (Participants) | 104 | 106 | 65 | 52
  Diarrhoea: Change at Cycle 8 Day 1 | 5.1 (19.6) | -0.9 (21.3) | 5.6 (20.9) | -3.2 (16.5)
  Diarrhoea: Change at Cycle 9 Day 1: number analyzed (Participants) | 100 | 101 | 62 | 52
  Diarrhoea: Change at Cycle 9 Day 1 | 7.7 (25.0) | 0.7 (24.5) | 4.3 (19.5) | -1.9 (23.3)
  Diarrhoea: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 62 | 47
  Diarrhoea: Change at Cycle 10 Day 1 | 6.9 (21.6) | -0.3 (22.3) | 5.9 (23.8) | -2.1 (18.9)
  Diarrhoea: Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 93 | 57 | 48
  Diarrhoea: Change at Cycle 11 Day 1 | 6.1 (19.6) | 1.1 (23.3) | 4.7 (23.1) | -0.7 (20.0)
  Diarrhoea: Change at Cycle 12 Day 1: number analyzed (Participants) | 90 | 91 | 55 | 47
  Diarrhoea: Change at Cycle 12 Day 1 | 7.4 (25.4) | -0.7 (23.3) | 7.9 (24.8) | -0.7 (19.0)
  Diarrhoea: Change at Cycle 13 Day 1: number analyzed (Participants) | 82 | 89 | 54 | 45
  Diarrhoea: Change at Cycle 13 Day 1 | 8.5 (24.5) | 0.4 (25.4) | 8.0 (28.9) | -1.5 (20.0)
  Diarrhoea: Change at End of Treatment: number analyzed (Participants) | 123 | 125 | 67 | 75
  Diarrhoea: Change at End of Treatment | 0.8 (21.5) | 0.0 (20.7) | -1.0 (16.4) | -1.8 (18.9)
  Diarrhoea: Change at PT 13 Weeks: number analyzed (Participants) | 90 | 74 | 56 | 38
  Diarrhoea: Change at PT 13 Weeks | -0.4 (15.4) | -1.8 (24.0) | 0.0 (18.0) | 0.0 (15.5)
  Diarrhoea: Change at PT 26 Weeks: number analyzed (Participants) | 89 | 72 | 47 | 35
  Diarrhoea: Change at PT 26 Weeks | -2.2 (16.5) | -3.2 (24.5) | 0.7 (8.5) | -1.9 (19.7)
  Diarrhoea: Change at PT 39 Weeks: number analyzed (Participants) | 79 | 68 | 41 | 33
  Diarrhoea: Change at PT 39 Weeks | -1.7 (15.9) | -4.9 (23.2) | 1.6 (14.8) | 0.0 (18.6)
  Diarrhoea: Change at PT 52 Weeks: number analyzed (Participants) | 75 | 62 | 27 | 25
  Diarrhoea: Change at PT 52 Weeks | -1.8 (17.2) | -3.8 (23.5) | -1.2 (21.6) | 0.0 (19.2)
  Diarrhoea: Change at PT 65 Weeks: number analyzed (Participants) | 53 | 38 | 17 | 18
  Diarrhoea: Change at PT 65 Weeks | 0.0 (19.6) | -6.1 (29.9) | 2.0 (8.1) | -7.4 (24.4)
  Diarrhoea: Change at PT 78 Weeks: number analyzed (Participants) | 46 | 33 | 15 | 9
  Diarrhoea: Change at PT 78 Weeks | -0.7 (20.5) | -7.1 (29.8) | 0.0 (0.0) | -3.7 (11.1)
  Diarrhoea: Change at PT 91 Weeks: number analyzed (Participants) | 33 | 29 | 15 | 12
  Diarrhoea: Change at PT 91 Weeks | 4.0 (16.2) | -9.2 (25.0) | 0.0 (0.0) | -8.3 (28.9)
  Diarrhoea: Change at PT 104 Weeks: number analyzed (Participants) | 27 | 25 | 10 | 9
  Diarrhoea: Change at PT 104 Weeks | 0.0 (9.2) | -5.3 (28.3) | 3.3 (10.5) | -11.1 (33.3)
  Diarrhoea: Change at PT 117 Weeks: number analyzed (Participants) | 22 | 17 | 8 | 5
  Diarrhoea: Change at PT 117 Weeks | 0.0 (10.3) | -11.8 (31.0) | 0.0 (0.0) | 0.0 (0.0)
  Diarrhoea: Change at PT 130 Weeks: number analyzed (Participants) | 17 | 12 | 5 | 5
  Diarrhoea: Change at PT 130 Weeks | -2.0 (8.1) | -2.8 (43.7) | 6.7 (14.9) | 13.3 (18.3)
  Diarrhoea: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Diarrhoea: Change at PT 143 Weeks | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Diarrhoea: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Diarrhoea: Change at PT 156 Weeks | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  | 0.0 (0.0)
  Diarrhoea: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Diarrhoea: Change at PT 169 Weeks | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Diarrhoea: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Diarrhoea: Change at PT 182 Weeks | 0.0 (0.0) |  |  |
  Diarrhoea: Change at PT/Discontinuation: number analyzed (Participants) | 8 | 1 | 6 | 1
  Diarrhoea: Change at PT/Discontinuation | 0.0 (17.8) | -33.3 (NA) — 1 participant was analyzed, so standard deviation is not applicable. | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable.
  Dyspnoea: Cycle 1 Day 1 (Baseline) | 3.6 (10.4) | 4.8 (12.9) | 5.0 (12.0) | 3.0 (10.8)
  Dyspnoea: Change at Cycle 1 Day 8: number analyzed (Participants) | 24 | 22 | 16 | 19
  Dyspnoea: Change at Cycle 1 Day 8 | 4.2 (11.3) | -1.5 (7.1) | 4.2 (16.7) | -1.8 (7.6)
  Dyspnoea: Change at Cycle 1 Day 15: number analyzed (Participants) | 132 | 139 | 80 | 84
  Dyspnoea: Change at Cycle 1 Day 15 | 6.3 (18.9) | 0.2 (8.5) | 2.9 (15.2) | 1.2 (12.1)
  Dyspnoea: Change at Cycle 1 Day 22: number analyzed (Participants) | 21 | 21 | 15 | 17
  Dyspnoea: Change at Cycle 1 Day 22 | 4.8 (12.0) | -1.6 (7.3) | 0.0 (17.8) | 0.0 (0.0)
  Dyspnoea: Change at Cycle 2 Day 1: number analyzed (Participants) | 126 | 142 | 83 | 84
  Dyspnoea: Change at Cycle 2 Day 1 | 1.9 (13.5) | 0.2 (11.6) | 4.8 (20.9) | 3.2 (14.3)
  Dyspnoea: Change at Cycle 2 Day 15: number analyzed (Participants) | 119 | 134 | 80 | 81
  Dyspnoea: Change at Cycle 2 Day 15 | 2.8 (16.0) | 1.0 (13.5) | 4.6 (18.9) | 4.1 (17.0)
  Dyspnoea: Change at Cycle 3 Day 1: number analyzed (Participants) | 119 | 129 | 81 | 78
  Dyspnoea: Change at Cycle 3 Day 1 | 3.4 (17.0) | 1.8 (13.4) | 3.7 (18.3) | 3.8 (12.0)
  Dyspnoea: Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 129 | 78 | 76
  Dyspnoea: Change at Cycle 4 Day 1 | 3.1 (15.6) | 3.1 (14.7) | 3.0 (18.8) | 1.8 (14.3)
  Dyspnoea: Change at Cycle 5 Day 1: number analyzed (Participants) | 110 | 116 | 72 | 64
  Dyspnoea: Change at Cycle 5 Day 1 | 5.2 (14.4) | 4.0 (14.7) | 3.7 (19.0) | 3.1 (15.4)
  Dyspnoea: Change at Cycle 6 Day 1: number analyzed (Participants) | 106 | 112 | 69 | 63
  Dyspnoea: Change at Cycle 6 Day 1 | 3.8 (16.8) | 2.4 (13.9) | 3.9 (19.4) | 2.1 (15.7)
  Dyspnoea: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 108 | 68 | 59
  Dyspnoea: Change at Cycle 7 Day 1 | 5.3 (16.7) | 3.7 (17.3) | 3.9 (17.8) | 2.8 (12.8)
  Dyspnoea: Change at Cycle 8 Day 1: number analyzed (Participants) | 104 | 106 | 65 | 53
  Dyspnoea: Change at Cycle 8 Day 1 | 4.2 (16.5) | 4.1 (17.6) | 2.6 (14.8) | 3.1 (13.5)
  Dyspnoea: Change at Cycle 9 Day 1: number analyzed (Participants) | 100 | 101 | 63 | 52
  Dyspnoea: Change at Cycle 9 Day 1 | 5.7 (17.1) | 5.3 (16.8) | 2.1 (16.8) | 4.5 (18.7)
  Dyspnoea: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 63 | 47
  Dyspnoea: Change at Cycle 10 Day 1 | 5.2 (20.1) | 4.5 (16.4) | 6.3 (18.8) | 3.5 (12.5)
  Dyspnoea: Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 93 | 57 | 48
  Dyspnoea: Change at Cycle 11 Day 1 | 5.7 (19.4) | 5.0 (19.0) | 7.0 (20.6) | 3.5 (14.2)
  Dyspnoea: Change at Cycle 12 Day 1: number analyzed (Participants) | 90 | 91 | 55 | 48
  Dyspnoea: Change at Cycle 12 Day 1 | 6.7 (24.1) | 5.5 (18.1) | 3.6 (18.9) | 5.6 (15.9)
  Dyspnoea: Change at Cycle 13 Day 1: number analyzed (Participants) | 82 | 89 | 54 | 45
  Dyspnoea: Change at Cycle 13 Day 1 | 6.5 (19.2) | 4.9 (15.5) | 4.9 (19.9) | 5.9 (14.7)
  Dyspnoea: Change at End of Treatment: number analyzed (Participants) | 123 | 125 | 67 | 75
  Dyspnoea: Change at End of Treatment | 4.1 (14.5) | 2.4 (19.9) | 3.0 (18.1) | 6.2 (16.2)
  Dyspnoea: Change at PT 13 Weeks: number analyzed (Participants) | 90 | 74 | 55 | 38
  Dyspnoea: Change at PT 13 Weeks | 3.0 (17.1) | 3.2 (16.7) | 3.0 (16.1) | 2.6 (12.0)
  Dyspnoea: Change at PT 26 Weeks: number analyzed (Participants) | 90 | 72 | 47 | 35
  Dyspnoea: Change at PT 26 Weeks | 4.8 (16.2) | 1.4 (16.3) | 3.5 (19.9) | -1.0 (5.6)
  Dyspnoea: Change at PT 39 Weeks: number analyzed (Participants) | 79 | 68 | 42 | 33
  Dyspnoea: Change at PT 39 Weeks | 1.7 (14.0) | 2.5 (13.3) | 4.8 (18.9) | 3.0 (12.8)
  Dyspnoea: Change at PT 52 Weeks: number analyzed (Participants) | 76 | 62 | 27 | 25
  Dyspnoea: Change at PT 52 Weeks | 1.8 (15.3) | 3.8 (16.1) | 2.5 (15.8) | 5.3 (15.8)
  Dyspnoea: Change at PT 65 Weeks: number analyzed (Participants) | 53 | 38 | 17 | 18
  Dyspnoea: Change at PT 65 Weeks | 3.8 (14.1) | 6.1 (15.2) | -3.9 (11.1) | 1.9 (7.9)
  Dyspnoea: Change at PT 78 Weeks: number analyzed (Participants) | 46 | 33 | 15 | 9
  Dyspnoea: Change at PT 78 Weeks | 4.3 (13.3) | 7.1 (18.2) | 0.0 (21.8) | 0.0 (16.7)
  Dyspnoea: Change at PT 91 Weeks: number analyzed (Participants) | 33 | 29 | 15 | 12
  Dyspnoea: Change at PT 91 Weeks | 3.0 (9.7) | 5.7 (12.8) | -2.2 (15.3) | 0.0 (14.2)
  Dyspnoea: Change at PT 104 Weeks: number analyzed (Participants) | 27 | 25 | 10 | 8
  Dyspnoea: Change at PT 104 Weeks | 0.0 (16.0) | 6.7 (16.7) | 0.0 (22.2) | 8.3 (15.4)
  Dyspnoea: Change at PT 117 Weeks: number analyzed (Participants) | 22 | 17 | 9 | 5
  Dyspnoea: Change at PT 117 Weeks | 0.0 (14.5) | 5.9 (13.1) | -3.7 (20.0) | 6.7 (14.9)
  Dyspnoea: Change at PT 130 Weeks: number analyzed (Participants) | 17 | 12 | 5 | 5
  Dyspnoea: Change at PT 130 Weeks | -2.0 (8.1) | 0.0 (0.0) | 0.0 (23.6) | 13.3 (18.3)
  Dyspnoea: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Dyspnoea: Change at PT 143 Weeks | 9.5 (25.2) | 0.0 (0.0) | -11.1 (19.2) | 0.0 (0.0)
  Dyspnoea: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Dyspnoea: Change at PT 156 Weeks | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  | 16.7 (23.6)
  Dyspnoea: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Dyspnoea: Change at PT 169 Weeks | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Dyspnoea: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Dyspnoea: Change at PT 182 Weeks | 0.0 (0.0) |  |  |
  Dyspnoea: Change at PT/Discontinuation: number analyzed (Participants) | 8 | 1 | 6 | 1
  Dyspnoea: Change at PT/Discontinuation | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable
  Emotional functioning: Cycle 1 Day 1 (Baseline) | 83.8 (15.1) | 86.1 (16.4) | 81.6 (21.5) | 84.5 (17.4)
  Emotional functioning: Change at Cycle 1 Day 8: number analyzed (Participants) | 24 | 22 | 16 | 19
  Emotional functioning: Change at Cycle 1 Day 8 | -4.5 (15.5) | 1.9 (12.0) | 3.6 (11.4) | 1.8 (14.0)
  Emotional functioning: Change at Cycle 1 Day 15: number analyzed (Participants) | 132 | 139 | 78 | 84
  Emotional functioning: Change at Cycle 1 Day 15 | -5.2 (18.0) | 1.9 (12.3) | -1.0 (16.6) | 3.8 (12.0)
  Emotional functioning: Change at Cycle 1 Day 22: number analyzed (Participants) | 22 | 21 | 15 | 17
  Emotional functioning: Change at Cycle 1 Day 22 | -6.4 (20.6) | 2.4 (9.9) | -0.6 (12.8) | -0.5 (17.3)
  Emotional functioning: Change at Cycle 2 Day 1: number analyzed (Participants) | 127 | 142 | 82 | 84
  Emotional functioning: Change at Cycle 2 Day 1 | -1.2 (16.0) | 2.5 (13.2) | -1.0 (17.5) | 4.0 (12.7)
  Emotional functioning: Change at Cycle 2 Day 15: number analyzed (Participants) | 119 | 134 | 80 | 80
  Emotional functioning: Change at Cycle 2 Day 15 | 0.2 (18.7) | 2.0 (15.4) | -0.5 (11.7) | 3.8 (13.6)
  Emotional functioning: Change at Cycle 3 Day 1: number analyzed (Participants) | 119 | 129 | 81 | 78
  Emotional functioning: Change at Cycle 3 Day 1 | -0.1 (17.3) | 2.3 (13.2) | -0.8 (16.8) | 3.5 (13.9)
  Emotional functioning: Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 129 | 78 | 76
  Emotional functioning: Change at Cycle 4 Day 1 | -2.7 (18.9) | 1.8 (15.1) | -1.2 (15.9) | 2.4 (14.9)
  Emotional functioning: Change at Cycle 5 Day 1: number analyzed (Participants) | 110 | 116 | 72 | 64
  Emotional functioning: Change at Cycle 5 Day 1 | -3.5 (19.8) | -0.2 (18.4) | -0.8 (15.4) | 3.0 (14.4)
  Emotional functioning: Change at Cycle 6 Day 1: number analyzed (Participants) | 106 | 112 | 69 | 63
  Emotional functioning: Change at Cycle 6 Day 1 | -2.8 (17.5) | -0.7 (16.7) | -2.6 (16.0) | 1.4 (18.7)
  Emotional functioning: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 108 | 68 | 59
  Emotional functioning: Change at Cycle 7 Day 1 | -3.0 (18.5) | 0.5 (16.4) | -2.3 (16.1) | -0.5 (14.4)
  Emotional functioning: Change at Cycle 8 Day 1: number analyzed (Participants) | 104 | 106 | 65 | 53
  Emotional functioning: Change at Cycle 8 Day 1 | -3.5 (20.0) | -0.9 (15.5) | -1.9 (15.9) | 0.2 (13.1)
  Emotional functioning: Change at Cycle 9 Day 1: number analyzed (Participants) | 100 | 101 | 63 | 52
  Emotional functioning: Change at Cycle 9 Day 1 | -1.6 (22.1) | -0.9 (17.0) | 0.1 (15.8) | -0.2 (16.1)
  Emotional functioning: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 63 | 47
  Emotional functioning: Change at Cycle 10 Day 1 | -1.0 (20.5) | -1.1 (14.3) | -0.1 (16.5) | 0.0 (14.6)
  Emotional functioning: Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 93 | 57 | 48
  Emotional functioning: Change at Cycle 11 Day 1 | 0.0 (19.6) | 0.5 (14.1) | 1.2 (15.7) | 0.7 (14.3)
  Emotional functioning: Change at Cycle 12 Day 1: number analyzed (Participants) | 90 | 91 | 55 | 48
  Emotional functioning: Change at Cycle 12 Day 1 | -2.3 (20.0) | -2.2 (16.4) | 1.1 (14.6) | -1.6 (14.1)
  Emotional functioning: Change at Cycle 13 Day 1: number analyzed (Participants) | 82 | 89 | 54 | 45
  Emotional functioning: Change at Cycle 13 Day 1 | -2.0 (20.4) | -2.5 (18.6) | 0.2 (16.5) | 0.2 (13.5)
  Emotional functioning: Change at End of Treatment: number analyzed (Participants) | 123 | 125 | 67 | 75
  Emotional functioning: Change at End of Treatment | 1.5 (18.8) | -2.0 (19.6) | 2.2 (22.2) | -4.4 (19.9)
  Emotional functioning: Change at PT 13 Weeks: number analyzed (Participants) | 90 | 74 | 56 | 38
  Emotional functioning: Change at PT 13 Weeks | 3.2 (17.4) | -1.0 (19.5) | 6.4 (16.7) | 3.5 (13.8)
  Emotional functioning: Change at PT 26 Weeks: number analyzed (Participants) | 90 | 72 | 47 | 35
  Emotional functioning: Change at PT 26 Weeks | 4.9 (18.3) | -1.4 (14.1) | 3.0 (18.2) | 1.2 (16.2)
  Emotional functioning: Change at PT 39 Weeks: number analyzed (Participants) | 79 | 68 | 41 | 33
  Emotional functioning: Change at PT 39 Weeks | 2.5 (15.5) | -0.2 (14.9) | 4.1 (19.0) | 2.3 (12.9)
  Emotional functioning: Change at PT 52 Weeks: number analyzed (Participants) | 76 | 62 | 27 | 25
  Emotional functioning: Change at PT 52 Weeks | 2.4 (17.8) | -0.7 (16.3) | 9.0 (16.8) | 1.7 (14.2)
  Emotional functioning: Change at PT 65 Weeks: number analyzed (Participants) | 53 | 38 | 17 | 18
  Emotional functioning: Change at PT 65 Weeks | 1.1 (17.9) | -2.0 (17.5) | 10.3 (17.1) | 3.7 (16.0)
  Emotional functioning: Change at PT 78 Weeks: number analyzed (Participants) | 46 | 33 | 15 | 9
  Emotional functioning: Change at PT 78 Weeks | 2.9 (14.6) | -1.8 (22.1) | 8.9 (16.2) | 1.9 (10.8)
  Emotional functioning: Change at PT 91 Weeks: number analyzed (Participants) | 33 | 29 | 15 | 12
  Emotional functioning: Change at PT 91 Weeks | 1.8 (16.8) | 0.0 (17.3) | 13.3 (16.6) | -0.7 (20.6)
  Emotional functioning: Change at PT 104 Weeks: number analyzed (Participants) | 27 | 25 | 10 | 9
  Emotional functioning: Change at PT 104 Weeks | 6.5 (14.3) | -7.0 (21.9) | 4.2 (13.2) | 1.9 (20.7)
  Emotional functioning: Change at PT 117 Weeks: number analyzed (Participants) | 22 | 17 | 8 | 5
  Emotional functioning: Change at PT 117 Weeks | 7.2 (12.7) | -2.9 (14.7) | 0.0 (16.7) | 3.3 (29.8)
  Emotional functioning: Change at PT 130 Weeks: number analyzed (Participants) | 17 | 12 | 5 | 5
  Emotional functioning: Change at PT 130 Weeks | 8.7 (12.8) | -4.9 (15.3) | 3.3 (20.1) | 1.7 (32.5)
  Emotional functioning: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Emotional functioning: Change at PT 143 Weeks | 0.0 (18.0) | -4.2 (5.9) | 0.0 (25.0) | -16.7 (23.6)
  Emotional functioning: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Emotional functioning: Change at PT 156 Weeks | 22.2 (9.6) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable |  | 4.2 (53.0)
  Emotional functioning: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Emotional functioning: Change at PT 169 Weeks | 25.0 (11.8) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Emotional functioning: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Emotional functioning: Change at PT 182 Weeks | 16.7 (16.7) |  |  |
  Emotional functioning: Change at PT/Discont.: number analyzed (Participants) | 8 | 1 | 6 | 1
  Emotional functioning: Change at PT/Discont. | -5.2 (28.1) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. | 1.4 (11.1) | 8.3 (NA) — 1 participant was analyzed, so standard deviation is not applicable.
  Fatigue: Cycle 1 Day 1 (Baseline) | 13.2 (14.7) | 16.1 (19.4) | 15.5 (18.2) | 14.7 (18.6)
  Fatigue: Change at Cycle 1 Day 8: number analyzed (Participants) | 24 | 22 | 16 | 19
  Fatigue: Change at Cycle 1 Day 8 | 7.9 (19.0) | -0.3 (9.8) | 7.6 (13.3) | 5.3 (10.1)
  Fatigue: Change at Cycle 1 Day 15: number analyzed (Participants) | 132 | 139 | 80 | 84
  Fatigue: Change at Cycle 1 Day 15 | 22.6 (26.1) | 2.3 (14.2) | 18.2 (27.0) | 3.4 (13.1)
  Fatigue: Change at Cycle 1 Day 22: number analyzed (Participants) | 22 | 21 | 15 | 17
  Fatigue: Change at Cycle 1 Day 22 | 15.2 (21.3) | -1.9 (14.4) | 17.0 (21.4) | 9.2 (15.8)
  Fatigue: Change at Cycle 2 Day 1: number analyzed (Participants) | 127 | 142 | 83 | 84
  Fatigue: Change at Cycle 2 Day 1 | 13.2 (22.0) | 2.5 (15.2) | 13.7 (24.2) | 2.5 (14.5)
  Fatigue: Change at Cycle 2 Day 15: number analyzed (Participants) | 119 | 134 | 80 | 81
  Fatigue: Change at Cycle 2 Day 15 | 15.2 (23.5) | 1.5 (18.2) | 10.7 (19.9) | 2.1 (16.5)
  Fatigue: Change at Cycle 3 Day 1: number analyzed (Participants) | 119 | 129 | 81 | 78
  Fatigue: Change at Cycle 3 Day 1 | 14.1 (22.5) | 1.5 (16.4) | 12.6 (23.1) | 4.7 (15.9)
  Fatigue: Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 129 | 78 | 76
  Fatigue: Change at Cycle 4 Day 1 | 12.6 (21.7) | 2.0 (18.4) | 13.3 (23.1) | 3.2 (18.1)
  Fatigue: Change at Cycle 5 Day 1: number analyzed (Participants) | 110 | 117 | 72 | 64
  Fatigue: Change at Cycle 5 Day 1 | 14.2 (23.7) | 1.9 (16.1) | 13.6 (18.9) | 4.7 (17.2)
  Fatigue: Change at Cycle 6 Day 1: number analyzed (Participants) | 106 | 112 | 69 | 63
  Fatigue: Change at Cycle 6 Day 1 | 11.9 (21.6) | 1.5 (17.4) | 13.8 (22.2) | 3.0 (18.7)
  Fatigue: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 108 | 68 | 59
  Fatigue: Change at Cycle 7 Day 1 | 13.1 (21.0) | 0.2 (18.3) | 13.2 (23.2) | 6.0 (17.7)
  Fatigue: Change at Cycle 8 Day 1: number analyzed (Participants) | 105 | 106 | 65 | 53
  Fatigue: Change at Cycle 8 Day 1 | 14.1 (23.9) | 3.9 (21.9) | 12.7 (22.7) | 5.0 (15.5)
  Fatigue: Change at Cycle 9 Day 1: number analyzed (Participants) | 100 | 101 | 63 | 52
  Fatigue: Change at Cycle 9 Day 1 | 16.3 (25.3) | 2.7 (20.5) | 13.7 (24.1) | 6.0 (21.3)
  Fatigue: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 63 | 47
  Fatigue: Change at Cycle 10 Day 1 | 11.3 (22.6) | 3.4 (18.7) | 11.3 (25.0) | 3.3 (16.2)
  Fatigue: Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 93 | 57 | 48
  Fatigue: Change at Cycle 11 Day 1 | 11.5 (22.7) | 2.7 (18.2) | 10.7 (20.9) | 7.6 (18.4)
  Fatigue: Change at Cycle 12 Day 1: number analyzed (Participants) | 90 | 91 | 55 | 48
  Fatigue: Change at Cycle 12 Day 1 | 10.3 (23.8) | 2.1 (16.2) | 10.7 (22.5) | 3.2 (17.0)
  Fatigue: Change at Cycle 13 Day 1: number analyzed (Participants) | 82 | 89 | 54 | 45
  Fatigue: Change at Cycle 13 Day 1 | 11.1 (23.1) | 4.0 (19.0) | 13.4 (26.6) | 4.7 (15.6)
  Fatigue: Change at End of Treatment: number analyzed (Participants) | 123 | 125 | 67 | 75
  Fatigue: Change at End of Treatment | 6.5 (21.3) | 2.2 (24.2) | 3.3 (21.9) | 6.4 (20.9)
  Fatigue: Change at PT 13 Weeks: number analyzed (Participants) | 90 | 74 | 56 | 38
  Fatigue: Change at PT 13 Weeks | 1.6 (18.4) | 0.7 (19.8) | -1.2 (19.0) | 1.5 (14.9)
  Fatigue: Change at PT 26 Weeks: number analyzed (Participants) | 90 | 72 | 47 | 35
  Fatigue: Change at PT 26 Weeks | 2.5 (18.4) | 1.0 (15.5) | 0.5 (21.6) | -1.3 (18.8)
  Fatigue: Change at PT 39 Weeks: number analyzed (Participants) | 79 | 68 | 42 | 33
  Fatigue: Change at PT 39 Weeks | -1.0 (16.9) | 0.7 (17.2) | -0.5 (18.2) | -0.3 (12.6)
  Fatigue: Change at PT 52 Weeks: number analyzed (Participants) | 76 | 62 | 27 | 25
  Fatigue: Change at PT 52 Weeks | 1.6 (16.7) | 1.7 (17.6) | -1.2 (14.6) | 1.3 (20.6)
  Fatigue: Change at PT 65 Weeks: number analyzed (Participants) | 53 | 38 | 17 | 18
  Fatigue: Change at PT 65 Weeks | 1.3 (16.5) | 4.4 (18.5) | -4.6 (11.8) | -1.2 (17.8)
  Fatigue: Change at PT 78 Weeks: number analyzed (Participants) | 46 | 33 | 15 | 9
  Fatigue: Change at PT 78 Weeks | 2.4 (16.2) | 4.7 (20.8) | -4.4 (10.1) | -4.9 (18.5)
  Fatigue: Change at PT 91 Weeks: number analyzed (Participants) | 33 | 29 | 15 | 12
  Fatigue: Change at PT 91 Weeks | -0.8 (16.3) | 3.8 (18.8) | -3.7 (15.5) | -2.8 (26.0)
  Fatigue: Change at PT 104 Weeks: number analyzed (Participants) | 27 | 25 | 10 | 9
  Fatigue: Change at PT 104 Weeks | -1.2 (14.6) | 8.9 (18.7) | -1.1 (17.7) | -1.2 (29.1)
  Fatigue: Change at PT 117 Weeks: number analyzed (Participants) | 22 | 17 | 9 | 5
  Fatigue: Change at PT 117 Weeks | -3.0 (13.4) | 4.2 (19.2) | -7.4 (15.7) | 0.0 (28.3)
  Fatigue: Change at PT 130 Weeks: number analyzed (Participants) | 17 | 12 | 5 | 5
  Fatigue: Change at PT 130 Weeks | -0.7 (15.5) | 6.5 (19.2) | -4.4 (16.9) | 0.0 (33.3)
  Fatigue: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Fatigue: Change at PT 143 Weeks | -1.6 (14.9) | 5.6 (7.9) | -3.7 (17.0) | 16.7 (23.6)
  Fatigue: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Fatigue: Change at PT 156 Weeks | -11.1 (11.1) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  | 33.3 (15.7)
  Fatigue: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Fatigue: Change at PT 169 Weeks | -16.7 (7.9) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Fatigue: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Fatigue: Change at PT 182 Weeks | -14.8 (6.4) |  |  |
  Fatigue: Change at PT/Discontinuation: number analyzed (Participants) | 8 | 1 | 6 | 1
  Fatigue: Change at PT/Discontinuation | 6.9 (16.7) | -22.2 (NA) — 1 participant was analyzed, so standard deviation is not applicable. | -11.1 (25.3) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable.
  Financial difficulties: Cycle 1 Day 1 (Baseline): number analyzed (Participants) | 137 | 147 | 87 | 88
  Financial difficulties: Cycle 1 Day 1 (Baseline) | 12.4 (25.2) | 20.9 (30.0) | 16.5 (30.4) | 15.9 (26.3)
  Financial difficulties: Change at Cycle 1 Day 8: number analyzed (Participants) | 24 | 22 | 16 | 19
  Financial difficulties: Change at Cycle 1 Day 8 | -9.7 (25.0) | -3.0 (14.2) | 2.1 (8.3) | -7.0 (17.8)
  Financial difficulties: Change at Cycle 1 Day 15: number analyzed (Participants) | 131 | 139 | 78 | 84
  Financial difficulties: Change at Cycle 1 Day 15 | 1.5 (17.5) | -1.9 (20.0) | 0.0 (15.2) | -4.4 (21.2)
  Financial difficulties: Change at Cycle 1 Day 22: number analyzed (Participants) | 22 | 21 | 15 | 17
  Financial difficulties: Change at Cycle 1 Day 22 | -1.5 (26.2) | -3.2 (14.5) | 0.0 (0.0) | 0.0 (20.4)
  Financial difficulties: Change at Cycle 2 Day 1: number analyzed (Participants) | 126 | 141 | 82 | 83
  Financial difficulties: Change at Cycle 2 Day 1 | 0.0 (17.9) | -3.1 (21.0) | 0.8 (16.5) | -4.4 (19.3)
  Financial difficulties: Change at Cycle 2 Day 15: number analyzed (Participants) | 119 | 134 | 80 | 79
  Financial difficulties: Change at Cycle 2 Day 15 | 1.1 (20.8) | -2.2 (20.1) | -0.4 (17.2) | -7.2 (20.4)
  Financial difficulties: Change at Cycle 3 Day 1: number analyzed (Participants) | 119 | 129 | 80 | 77
  Financial difficulties: Change at Cycle 3 Day 1 | 0.3 (21.5) | -5.2 (24.1) | 1.3 (20.2) | -5.6 (19.8)
  Financial difficulties: Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 129 | 78 | 75
  Financial difficulties: Change at Cycle 4 Day 1 | -0.8 (23.6) | -2.8 (24.3) | -0.4 (19.7) | -5.8 (18.5)
  Financial difficulties: Change at Cycle 5 Day 1: number analyzed (Participants) | 110 | 116 | 72 | 64
  Financial difficulties: Change at Cycle 5 Day 1 | 1.2 (23.0) | -5.5 (26.7) | 2.3 (18.0) | -7.8 (23.6)
  Financial difficulties: Change at Cycle 6 Day 1: number analyzed (Participants) | 106 | 112 | 69 | 63
  Financial difficulties: Change at Cycle 6 Day 1 | -0.6 (22.5) | -7.4 (26.4) | 2.9 (20.4) | -5.8 (22.0)
  Financial difficulties: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 107 | 68 | 59
  Financial difficulties: Change at Cycle 7 Day 1 | 1.9 (26.8) | -5.6 (26.1) | 4.9 (27.2) | -5.6 (21.6)
  Financial difficulties: Change at Cycle 8 Day 1: number analyzed (Participants) | 104 | 106 | 65 | 53
  Financial difficulties: Change at Cycle 8 Day 1 | -0.6 (23.2) | -4.7 (27.0) | 4.1 (26.7) | -3.1 (20.9)
  Financial difficulties: Change at Cycle 9 Day 1: number analyzed (Participants) | 100 | 101 | 63 | 52
  Financial difficulties: Change at Cycle 9 Day 1 | 2.0 (24.1) | -8.9 (23.0) | 4.2 (23.6) | -5.8 (20.6)
  Financial difficulties: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 63 | 47
  Financial difficulties: Change at Cycle 10 Day 1 | 1.0 (23.4) | -8.6 (25.1) | 2.6 (22.6) | -6.4 (20.4)
  Financial difficulties: Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 93 | 57 | 48
  Financial difficulties: Change at Cycle 11 Day 1 | 1.4 (21.4) | -7.5 (21.5) | 0.6 (20.4) | -8.3 (22.3)
  Financial difficulties: Change at Cycle 12 Day 1: number analyzed (Participants) | 89 | 90 | 55 | 48
  Financial difficulties: Change at Cycle 12 Day 1 | -0.4 (24.4) | -6.3 (23.9) | 0.0 (26.4) | -6.3 (23.5)
  Financial difficulties: Change at Cycle 13 Day 1: number analyzed (Participants) | 82 | 89 | 54 | 45
  Financial difficulties: Change at Cycle 13 Day 1 | 1.2 (23.7) | -6.0 (22.2) | -1.9 (27.8) | -8.1 (24.8)
  Financial difficulties: Change at End of Treatment: number analyzed (Participants) | 122 | 125 | 67 | 75
  Financial difficulties: Change at End of Treatment | 2.5 (23.1) | -3.7 (26.5) | -2.5 (23.4) | -0.9 (23.9)
  Financial difficulties: Change at PT 13 Weeks: number analyzed (Participants) | 90 | 74 | 56 | 38
  Financial difficulties: Change at PT 13 Weeks | 0.4 (26.2) | -5.9 (24.3) | -10.1 (27.6) | -8.8 (25.3)
  Financial difficulties: Change at PT 26 Weeks: number analyzed (Participants) | 89 | 72 | 47 | 35
  Financial difficulties: Change at PT 26 Weeks | -3.0 (22.3) | -6.0 (18.8) | -5.7 (26.3) | -7.6 (25.7)
  Financial difficulties: Change at PT 39 Weeks: number analyzed (Participants) | 78 | 68 | 41 | 33
  Financial difficulties: Change at PT 39 Weeks | -1.7 (22.1) | -7.8 (25.8) | -2.4 (28.3) | -8.1 (26.4)
  Financial difficulties: Change at PT 52 Weeks: number analyzed (Participants) | 75 | 62 | 27 | 25
  Financial difficulties: Change at PT 52 Weeks | -2.2 (21.5) | -5.4 (21.1) | -11.1 (24.5) | -1.3 (32.6)
  Financial difficulties: Change at PT 65 Weeks: number analyzed (Participants) | 52 | 38 | 17 | 18
  Financial difficulties: Change at PT 65 Weeks | 2.6 (26.3) | -6.1 (30.9) | -9.8 (19.6) | -7.4 (31.4)
  Financial difficulties: Change at PT 78 Weeks: number analyzed (Participants) | 45 | 33 | 15 | 9
  Financial difficulties: Change at PT 78 Weeks | 2.2 (27.9) | -8.1 (31.2) | -11.1 (20.6) | 0.0 (16.7)
  Financial difficulties: Change at PT 91 Weeks: number analyzed (Participants) | 31 | 29 | 15 | 12
  Financial difficulties: Change at PT 91 Weeks | 0.0 (27.2) | -10.3 (29.7) | -11.1 (20.6) | -11.1 (32.8)
  Financial difficulties: Change at PT 104 Weeks: number analyzed (Participants) | 26 | 25 | 10 | 9
  Financial difficulties: Change at PT 104 Weeks | -2.6 (18.7) | -8.0 (30.9) | -13.3 (23.3) | -18.5 (37.7)
  Financial difficulties: Change at PT 117 Weeks: number analyzed (Participants) | 22 | 17 | 8 | 5
  Financial difficulties: Change at PT 117 Weeks | -6.1 (22.1) | -5.9 (24.3) | -4.2 (11.8) | -13.3 (18.3)
  Financial difficulties: Change at PT 130 Weeks: number analyzed (Participants) | 17 | 12 | 5 | 5
  Financial difficulties: Change at PT 130 Weeks | -7.8 (27.7) | -5.6 (31.2) | 0.0 (0.0) | -20.0 (29.8)
  Financial difficulties: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Financial difficulties: Change at PT 143 Weeks | 4.8 (40.5) | 16.7 (23.6) | 0.0 (0.0) | 0.0 (0.0)
  Financial difficulties: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Financial difficulties: Change at PT 156 Weeks | -22.2 (38.5) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  | -16.7 (23.6)
  Financial difficulties: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Financial difficulties: Change at PT 169 Weeks | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Financial difficulties: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Financial difficulties: Change at PT 182 Weeks | -22.2 (38.5) |  |  |
  Financial difficulties: Change at PT/Discontin.: number analyzed (Participants) | 8 | 1 | 6 | 1
  Financial difficulties: Change at PT/Discontin. | 0.0 (17.8) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable.
  Nausea and vomiting: Cycle 1 Day 1 (Baseline) | 1.4 (5.1) | 1.8 (9.6) | 1.9 (7.4) | 1.3 (5.2)
  Nausea and vomiting: Change at Cycle 1 Day 8: number analyzed (Participants) | 24 | 22 | 16 | 19
  Nausea and vomiting: Change at Cycle 1 Day 8 | 4.2 (8.9) | 0.8 (6.3) | 5.2 (8.0) | 3.5 (8.9)
  Nausea and vomiting: Change at Cycle 1 Day 15: number analyzed (Participants) | 132 | 139 | 80 | 84
  Nausea and vomiting: Change at Cycle 1 Day 15 | 9.8 (16.9) | 1.8 (6.9) | 8.8 (17.0) | 1.2 (7.7)
  Nausea and vomiting: Change at Cycle 1 Day 22: number analyzed (Participants) | 22 | 21 | 15 | 17
  Nausea and vomiting: Change at Cycle 1 Day 22 | 6.1 (12.1) | 0.8 (6.4) | 5.6 (10.3) | 2.9 (8.8)
  Nausea and vomiting: Change at Cycle 2 Day 1: number analyzed (Participants) | 127 | 142 | 83 | 84
  Nausea and vomiting: Change at Cycle 2 Day 1 | 5.2 (12.9) | 0.9 (5.9) | 4.6 (11.1) | 1.4 (7.9)
  Nausea and vomiting: Change at Cycle 2 Day 15: number analyzed (Participants) | 119 | 134 | 80 | 81
  Nausea and vomiting: Change at Cycle 2 Day 15 | 6.3 (14.1) | 1.1 (8.5) | 2.9 (9.1) | 1.6 (10.4)
  Nausea and vomiting: Change at Cycle 3 Day 1: number analyzed (Participants) | 119 | 129 | 81 | 78
  Nausea and vomiting: Change at Cycle 3 Day 1 | 5.7 (13.1) | 1.6 (7.3) | 4.5 (9.9) | 1.3 (8.4)
  Nausea and vomiting: Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 129 | 78 | 76
  Nausea and vomiting: Change at Cycle 4 Day 1 | 5.6 (13.6) | 1.9 (11.7) | 6.6 (14.3) | 1.3 (10.8)
  Nausea and vomiting: Change at Cycle 5 Day 1: number analyzed (Participants) | 110 | 117 | 72 | 64
  Nausea and vomiting: Change at Cycle 5 Day 1 | 7.3 (16.4) | 2.6 (9.2) | 5.1 (10.7) | -0.5 (7.8)
  Nausea and vomiting: Change at Cycle 6 Day 1: number analyzed (Participants) | 106 | 112 | 69 | 63
  Nausea and vomiting: Change at Cycle 6 Day 1 | 5.3 (13.1) | 2.4 (9.7) | 6.3 (12.2) | -0.5 (7.9)
  Nausea and vomiting: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 108 | 68 | 59
  Nausea and vomiting: Change at Cycle 7 Day 1 | 4.7 (11.7) | 2.0 (7.8) | 4.2 (11.3) | 0.6 (6.9)
  Nausea and vomiting: Change at Cycle 8 Day 1: number analyzed (Participants) | 105 | 106 | 65 | 53
  Nausea and vomiting: Change at Cycle 8 Day 1 | 4.6 (11.9) | 1.1 (9.0) | 5.9 (15.7) | 2.5 (12.4)
  Nausea and vomiting: Change at Cycle 9 Day 1: number analyzed (Participants) | 100 | 101 | 63 | 52
  Nausea and vomiting: Change at Cycle 9 Day 1 | 5.5 (15.7) | 2.5 (10.4) | 4.0 (10.2) | 0.3 (7.0)
  Nausea and vomiting: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 63 | 47
  Nausea and vomiting: Change at Cycle 10 Day 1 | 5.2 (13.1) | 0.9 (10.3) | 4.8 (10.6) | 0.4 (6.5)
  Nausea and vomiting: Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 93 | 57 | 48
  Nausea and vomiting: Change at Cycle 11 Day 1 | 3.4 (10.9) | 2.0 (8.5) | 3.2 (8.6) | -0.3 (5.4)
  Nausea and vomiting: Change at Cycle 12 Day 1: number analyzed (Participants) | 90 | 91 | 55 | 48
  Nausea and vomiting: Change at Cycle 12 Day 1 | 4.3 (12.6) | 1.3 (7.9) | 4.8 (10.5) | 3.5 (13.7)
  Nausea and vomiting: Change at Cycle 13 Day 1: number analyzed (Participants) | 82 | 89 | 54 | 45
  Nausea and vomiting: Change at Cycle 13 Day 1 | 2.8 (11.7) | 1.7 (7.1) | 3.4 (9.9) | 2.2 (9.8)
  Nausea and vomiting: Change at End of Treatment: number analyzed (Participants) | 123 | 125 | 67 | 75
  Nausea and vomiting: Change at End of Treatment | 0.9 (6.5) | 0.3 (12.5) | 1.5 (11.9) | 3.8 (13.9)
  Nausea and vomiting: Change at PT 13 Weeks: number analyzed (Participants) | 90 | 74 | 56 | 38
  Nausea and vomiting: Change at PT 13 Weeks | 0.2 (6.4) | 1.8 (8.5) | 0.6 (6.3) | 0.9 (6.7)
  Nausea and vomiting: Change at PT 26 Weeks: number analyzed (Participants) | 90 | 72 | 47 | 35
  Nausea and vomiting: Change at PT 26 Weeks | 2.2 (8.7) | 0.7 (15.7) | 0.7 (10.4) | -1.0 (3.9)
  Nausea and vomiting: Change at PT 39 Weeks: number analyzed (Participants) | 79 | 68 | 42 | 33
  Nausea and vomiting: Change at PT 39 Weeks | 0.2 (5.7) | 0.2 (6.1) | 1.6 (8.1) | 1.5 (6.4)
  Nausea and vomiting: Change at PT 52 Weeks: number analyzed (Participants) | 76 | 62 | 27 | 25
  Nausea and vomiting: Change at PT 52 Weeks | 0.9 (6.0) | 0.3 (4.8) | 0.0 (4.6) | 0.7 (3.3)
  Nausea and vomiting: Change at PT 65 Weeks: number analyzed (Participants) | 53 | 38 | 17 | 18
  Nausea and vomiting: Change at PT 65 Weeks | 0.0 (5.7) | 3.5 (12.9) | -1.0 (4.0) | 2.8 (8.6)
  Nausea and vomiting: Change at PT 78 Weeks: number analyzed (Participants) | 46 | 33 | 15 | 9
  Nausea and vomiting: Change at PT 78 Weeks | 0.4 (5.5) | 2.0 (11.6) | -1.1 (4.3) | 1.9 (5.6)
  Nausea and vomiting: Change at PT 91 Weeks: number analyzed (Participants) | 32 | 29 | 15 | 12
  Nausea and vomiting: Change at PT 91 Weeks | 1.6 (6.5) | 2.3 (8.6) | -1.1 (4.3) | 1.4 (4.8)
  Nausea and vomiting: Change at PT 104 Weeks: number analyzed (Participants) | 27 | 25 | 10 | 9
  Nausea and vomiting: Change at PT 104 Weeks | 1.9 (10.7) | 0.0 (4.8) | 0.0 (0.0) | 0.0 (0.0)
  Nausea and vomiting: Change at PT 117 Weeks: number analyzed (Participants) | 22 | 17 | 9 | 5
  Nausea and vomiting: Change at PT 117 Weeks | -1.5 (4.9) | 4.9 (9.8) | -1.9 (5.6) | 0.0 (0.0)
  Nausea and vomiting: Change at PT 130 Weeks: number analyzed (Participants) | 17 | 12 | 5 | 5
  Nausea and vomiting: Change at PT 130 Weeks | 0.0 (5.9) | 4.2 (10.4) | -3.3 (7.5) | 0.0 (0.0)
  Nausea and vomiting: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Nausea and vomiting: Change at PT 143 Weeks | -2.4 (6.3) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Nausea and vomiting: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Nausea and vomiting: Change at PT 156 Weeks | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  | 8.3 (11.8)
  Nausea and vomiting: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Nausea and vomiting: Change at PT 169 Weeks | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Nausea and vomiting: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Nausea and vomiting: Change at PT 182 Weeks | 0.0 (0.0) |  |  |
  Nausea and vomiting: Change at PT/Discont.: number analyzed (Participants) | 8 | 1 | 6 | 1
  Nausea and vomiting: Change at PT/Discont. | 4.2 (11.8) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. | 8.3 (13.9) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable.
  Pain: Cycle 1 Day 1 (Baseline) | 11.6 (17.5) | 12.8 (21.6) | 10.9 (19.0) | 14.6 (23.9)
  Pain: Change at Cycle 1 Day 8: number analyzed (Participants) | 24 | 22 | 16 | 19
  Pain: Change at Cycle 1 Day 8 | 9.7 (22.5) | -1.5 (15.4) | 10.4 (14.8) | -3.5 (8.9)
  Pain: Change at Cycle 1 Day 15: number analyzed (Participants) | 132 | 139 | 80 | 84
  Pain: Change at Cycle 1 Day 15 | 20.8 (28.5) | 0.5 (12.4) | 16.3 (28.1) | -1.4 (14.7)
  Pain: Change at Cycle 1 Day 22: number analyzed (Participants) | 22 | 21 | 15 | 17
  Pain: Change at Cycle 1 Day 22 | 15.9 (28.9) | -3.2 (13.6) | 22.2 (18.5) | 9.8 (21.3)
  Pain: Change at Cycle 2 Day 1: number analyzed (Participants) | 127 | 142 | 83 | 84
  Pain: Change at Cycle 2 Day 1 | 12.9 (26.5) | 0.5 (15.1) | 15.1 (28.9) | -3.8 (18.0)
  Pain: Change at Cycle 2 Day 15: number analyzed (Participants) | 119 | 134 | 80 | 81
  Pain: Change at Cycle 2 Day 15 | 14.3 (27.5) | 2.4 (17.2) | 12.7 (23.3) | -3.5 (18.0)
  Pain: Change at Cycle 3 Day 1: number analyzed (Participants) | 119 | 129 | 81 | 78
  Pain: Change at Cycle 3 Day 1 | 11.8 (20.2) | 1.2 (16.3) | 13.2 (25.6) | -0.6 (17.1)
  Pain: Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 129 | 78 | 76
  Pain: Change at Cycle 4 Day 1 | 9.0 (22.1) | 4.0 (19.7) | 12.0 (25.9) | -2.4 (19.6)
  Pain: Change at Cycle 5 Day 1: number analyzed (Participants) | 110 | 117 | 72 | 64
  Pain: Change at Cycle 5 Day 1 | 12.7 (24.3) | 1.9 (17.6) | 14.6 (21.1) | -4.9 (20.5)
  Pain: Change at Cycle 6 Day 1: number analyzed (Participants) | 106 | 112 | 69 | 63
  Pain: Change at Cycle 6 Day 1 | 8.8 (22.7) | 2.2 (18.9) | 14.5 (22.9) | -3.7 (20.0)
  Pain: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 108 | 68 | 59
  Pain: Change at Cycle 7 Day 1 | 8.2 (21.4) | 0.9 (16.6) | 8.3 (20.5) | -2.0 (19.1)
  Pain: Change at Cycle 8 Day 1: number analyzed (Participants) | 105 | 106 | 65 | 53
  Pain: Change at Cycle 8 Day 1 | 11.0 (24.9) | 3.6 (20.1) | 12.1 (23.7) | -1.6 (18.3)
  Pain: Change at Cycle 9 Day 1: number analyzed (Participants) | 100 | 101 | 63 | 52
  Pain: Change at Cycle 9 Day 1 | 12.8 (27.5) | 3.6 (21.2) | 10.3 (23.5) | -0.3 (23.9)
  Pain: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 63 | 47
  Pain: Change at Cycle 10 Day 1 | 8.9 (22.0) | 1.9 (17.5) | 11.6 (24.6) | -3.2 (16.9)
  Pain: Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 93 | 57 | 48
  Pain: Change at Cycle 11 Day 1 | 10.0 (25.0) | 2.7 (21.3) | 13.5 (26.1) | -0.7 (24.3)
  Pain: Change at Cycle 12 Day 1: number analyzed (Participants) | 90 | 91 | 55 | 48
  Pain: Change at Cycle 12 Day 1 | 12.2 (24.6) | 1.3 (19.8) | 12.7 (19.5) | -2.1 (20.2)
  Pain: Change at Cycle 13 Day 1: number analyzed (Participants) | 82 | 89 | 54 | 45
  Pain: Change at Cycle 13 Day 1 | 11.6 (23.5) | 3.4 (21.2) | 16.4 (27.4) | -1.9 (22.0)
  Pain: Change at End of Treatment: number analyzed (Participants) | 123 | 125 | 67 | 75
  Pain: Change at End of Treatment | 4.9 (23.4) | 4.1 (23.3) | 6.7 (21.1) | 1.6 (21.4)
  Pain: Change at PT 13 Weeks: number analyzed (Participants) | 90 | 74 | 56 | 38
  Pain: Change at PT 13 Weeks | -0.6 (17.6) | -0.2 (18.2) | 4.2 (19.7) | -4.8 (23.5)
  Pain: Change at PT 26 Weeks: number analyzed (Participants) | 90 | 72 | 47 | 35
  Pain: Change at PT 26 Weeks | 1.1 (21.8) | -1.2 (16.6) | 7.1 (24.0) | -4.3 (19.5)
  Pain: Change at PT 39 Weeks: number analyzed (Participants) | 79 | 68 | 42 | 33
  Pain: Change at PT 39 Weeks | 0.6 (19.9) | 2.2 (22.1) | 7.5 (23.0) | -7.6 (23.2)
  Pain: Change at PT 52 Weeks: number analyzed (Participants) | 76 | 62 | 27 | 25
  Pain: Change at PT 52 Weeks | 2.0 (18.0) | 0.0 (16.3) | 9.3 (21.8) | -1.3 (20.4)
  Pain: Change at PT 65 Weeks: number analyzed (Participants) | 53 | 38 | 17 | 18
  Pain: Change at PT 65 Weeks | -0.3 (19.7) | 0.9 (21.2) | 6.9 (15.7) | -4.6 (12.5)
  Pain: Change at PT 78 Weeks: number analyzed (Participants) | 46 | 33 | 15 | 9
  Pain: Change at PT 78 Weeks | 0.7 (20.2) | 2.5 (19.6) | 1.1 (14.7) | -5.6 (8.3)
  Pain: Change at PT 91 Weeks: number analyzed (Participants) | 33 | 29 | 15 | 12
  Pain: Change at PT 91 Weeks | -2.5 (18.7) | 4.6 (25.9) | 4.4 (14.7) | -9.7 (21.9)
  Pain: Change at PT 104 Weeks: number analyzed (Participants) | 27 | 25 | 10 | 9
  Pain: Change at PT 104 Weeks | -1.2 (17.9) | 11.3 (22.4) | 3.3 (13.1) | -13.0 (21.7)
  Pain: Change at PT 117 Weeks: number analyzed (Participants) | 22 | 17 | 9 | 5
  Pain: Change at PT 117 Weeks | -4.5 (18.0) | 8.8 (22.9) | 1.9 (13.0) | -10.0 (25.3)
  Pain: Change at PT 130 Weeks: number analyzed (Participants) | 17 | 12 | 5 | 5
  Pain: Change at PT 130 Weeks | 2.9 (19.8) | 6.9 (31.3) | 6.7 (27.9) | -13.3 (32.1)
  Pain: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Pain: Change at PT 143 Weeks | -2.4 (20.2) | 8.3 (11.8) | 5.6 (25.5) | 0.0 (0.0)
  Pain: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Pain: Change at PT 156 Weeks | -22.2 (19.2) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  | 8.3 (11.8)
  Pain: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Pain: Change at PT 169 Weeks | -8.3 (11.8) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Pain: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Pain: Change at PT 182 Weeks | -22.2 (19.2) |  |  |
  Pain: Change at PT/Discontin.: number analyzed (Participants) | 8 | 1 | 6 | 1
  Pain: Change at PT/Discontin. | 12.5 (14.8) | -33.3 (NA) — 1 participant was analyzed, so standard deviation is not applicable. | -2.8 (19.5) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable.
  Physical functioning: Cycle 1 Day 1 (Baseline) | 92.7 (11.0) | 92.3 (11.6) | 91.3 (13.6) | 92.7 (13.1)
  Physical functioning: Change at Cycle 1 Day 8: number analyzed (Participants) | 24 | 22 | 16 | 19
  Physical functioning: Change at Cycle 1 Day 8 | -4.4 (8.7) | 0.3 (4.4) | -5.0 (6.7) | -2.5 (11.6)
  Physical functioning: Change at Cycle 1 Day 15: number analyzed (Participants) | 132 | 139 | 80 | 84
  Physical functioning: Change at Cycle 1 Day 15 | -9.7 (17.4) | -0.2 (8.2) | -7.4 (15.0) | -1.5 (6.5)
  Physical functioning: Change at Cycle 1 Day 22: number analyzed (Participants) | 22 | 21 | 15 | 17
  Physical functioning: Change at Cycle 1 Day 22 | -10.3 (16.6) | -0.6 (7.0) | -10.2 (15.3) | -2.7 (9.7)
  Physical functioning: Change at Cycle 2 Day 1: number analyzed (Participants) | 127 | 142 | 83 | 84
  Physical functioning: Change at Cycle 2 Day 1 | -6.2 (14.4) | -0.3 (9.1) | -9.2 (16.9) | -1.8 (8.2)
  Physical functioning: Change at Cycle 2 Day 15: number analyzed (Participants) | 119 | 134 | 80 | 81
  Physical functioning: Change at Cycle 2 Day 15 | -7.1 (16.4) | -0.7 (10.8) | -7.6 (13.9) | -1.4 (9.4)
  Physical functioning: Change at Cycle 3 Day 1: number analyzed (Participants) | 119 | 129 | 81 | 78
  Physical functioning: Change at Cycle 3 Day 1 | -6.6 (14.8) | -0.7 (11.0) | -7.3 (15.0) | -2.7 (10.4)
  Physical functioning: Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 129 | 78 | 76
  Physical functioning: Change at Cycle 4 Day 1 | -4.9 (13.1) | -0.2 (10.8) | -7.4 (13.8) | -1.0 (10.3)
  Physical functioning: Change at Cycle 5 Day 1: number analyzed (Participants) | 110 | 117 | 72 | 64
  Physical functioning: Change at Cycle 5 Day 1 | -6.1 (14.7) | -1.0 (11.3) | -5.6 (13.3) | -1.8 (12.7)
  Physical functioning: Change at Cycle 6 Day 1: number analyzed (Participants) | 106 | 112 | 69 | 63
  Physical functioning: Change at Cycle 6 Day 1 | -4.7 (14.5) | -0.8 (12.1) | -7.5 (15.2) | -0.6 (10.0)
  Physical functioning: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 108 | 68 | 59
  Physical functioning: Change at Cycle 7 Day 1 | -4.7 (13.6) | 0.4 (11.2) | -8.0 (12.7) | 0.2 (9.5)
  Physical functioning: Change at Cycle 8 Day 1: number analyzed (Participants) | 105 | 106 | 65 | 53
  Physical functioning: Change at Cycle 8 Day 1 | -5.2 (13.6) | -0.8 (13.1) | -6.7 (12.6) | -0.3 (11.0)
  Physical functioning: Change at Cycle 9 Day 1: number analyzed (Participants) | 100 | 101 | 63 | 52
  Physical functioning: Change at Cycle 9 Day 1 | -6.7 (18.2) | -0.5 (12.2) | -5.5 (10.6) | -1.5 (14.7)
  Physical functioning: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 63 | 47
  Physical functioning: Change at Cycle 10 Day 1 | -4.9 (14.0) | -1.6 (11.8) | -6.5 (13.2) | -1.7 (9.9)
  Physical functioning: Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 93 | 57 | 48
  Physical functioning: Change at Cycle 11 Day 1 | -4.2 (14.4) | -1.3 (10.8) | -6.0 (12.8) | -3.3 (13.5)
  Physical functioning: Change at Cycle 12 Day 1: number analyzed (Participants) | 90 | 91 | 55 | 48
  Physical functioning: Change at Cycle 12 Day 1 | -5.4 (15.7) | -1.6 (11.5) | -4.8 (11.9) | -0.6 (10.8)
  Physical functioning: Change at Cycle 13 Day 1: number analyzed (Participants) | 82 | 89 | 54 | 45
  Physical functioning: Change at Cycle 13 Day 1 | -4.5 (15.0) | -3.0 (14.7) | -5.6 (12.4) | -1.9 (12.3)
  Physical functioning: Change at End of Treatment: number analyzed (Participants) | 123 | 125 | 67 | 75
  Physical functioning: Change at End of Treatment | -2.8 (13.3) | -2.9 (16.0) | -5.8 (13.8) | -5.1 (14.7)
  Physical functioning: Change at PT 13 Weeks: number analyzed (Participants) | 90 | 74 | 56 | 38
  Physical functioning: Change at PT 13 Weeks | 0.5 (11.3) | 0.1 (9.8) | -0.8 (10.9) | -0.5 (12.6)
  Physical functioning: Change at PT 26 Weeks: number analyzed (Participants) | 90 | 72 | 47 | 35
  Physical functioning: Change at PT 26 Weeks | -1.9 (12.5) | 0.0 (8.5) | -4.1 (10.5) | 0.6 (12.6)
  Physical functioning: Change at PT 39 Weeks: number analyzed (Participants) | 79 | 68 | 42 | 33
  Physical functioning: Change at PT 39 Weeks | 0.4 (10.7) | -1.7 (13.5) | -3.3 (13.4) | 0.6 (8.1)
  Physical functioning: Change at PT 52 Weeks: number analyzed (Participants) | 76 | 62 | 27 | 25
  Physical functioning: Change at PT 52 Weeks | -1.4 (10.0) | -0.5 (11.7) | -1.4 (9.6) | -1.1 (14.2)
  Physical functioning: Change at PT 65 Weeks: number analyzed (Participants) | 53 | 38 | 17 | 18
  Physical functioning: Change at PT 65 Weeks | -0.9 (8.6) | -2.6 (13.6) | 2.7 (9.7) | -0.4 (10.3)
  Physical functioning: Change at PT 78 Weeks: number analyzed (Participants) | 46 | 33 | 15 | 9
  Physical functioning: Change at PT 78 Weeks | -0.5 (8.6) | -1.0 (10.8) | 2.7 (10.0) | -3.7 (11.6)
  Physical functioning: Change at PT 91 Weeks: number analyzed (Participants) | 33 | 29 | 15 | 12
  Physical functioning: Change at PT 91 Weeks | 0.2 (7.2) | -3.4 (12.9) | -0.9 (10.3) | 0.0 (17.5)
  Physical functioning: Change at PT 104 Weeks: number analyzed (Participants) | 27 | 25 | 10 | 9
  Physical functioning: Change at PT 104 Weeks | 2.5 (8.3) | -4.9 (10.3) | 1.3 (11.2) | 1.5 (18.2)
  Physical functioning: Change at PT 117 Weeks: number analyzed (Participants) | 22 | 17 | 9 | 5
  Physical functioning: Change at PT 117 Weeks | 1.2 (8.1) | -7.1 (14.2) | 0.7 (13.1) | 2.7 (19.2)
  Physical functioning: Change at PT 130 Weeks: number analyzed (Participants) | 17 | 12 | 5 | 5
  Physical functioning: Change at PT 130 Weeks | -1.2 (4.2) | -5.0 (11.4) | -2.7 (10.1) | 5.3 (20.2)
  Physical functioning: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Physical functioning: Change at PT 143 Weeks | 0.0 (8.6) | 0.0 (0.0) | -4.4 (20.4) | -3.3 (4.7)
  Physical functioning: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Physical functioning: Change at PT 156 Weeks | 2.2 (3.8) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  | -6.7 (9.4)
  Physical functioning: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Physical functioning: Change at PT 169 Weeks | 3.3 (4.7) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Physical functioning: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Physical functioning: Change at PT 182 Weeks | 2.2 (3.8) |  |  |
  Physical functioning: Change at PT/Discontin.: number analyzed (Participants) | 8 | 1 | 6 | 1
  Physical functioning: Change at PT/Discontin. | -0.8 (8.3) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable | 10.0 (15.6) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable.
  Global health status/QoL: Cycle 1 Day 1 (Baseline) | 79.0 (16.7) | 77.9 (18.4) | 76.5 (20.6) | 78.8 (17.6)
  Global health status/QoL: Change at Cycle 1 Day 8: number analyzed (Participants) | 24 | 22 | 16 | 19
  Global health status/QoL: Change at Cycle 1 Day 8 | -9.4 (20.5) | 0.4 (7.5) | -9.9 (15.9) | 1.3 (6.4)
  Global health status/QoL: Change at Cycle 1 Day 15: number analyzed (Participants) | 132 | 139 | 78 | 83
  Global health status/QoL: Change at Cycle 1 Day 15 | -19.1 (24.2) | -0.4 (11.4) | -14.5 (20.4) | -0.3 (11.7)
  Global health status/QoL: Change at Cycle 1 Day 22: number analyzed (Participants) | 22 | 21 | 15 | 17
  Global health status/QoL: Change at Cycle 1 Day 22 | -17.8 (27.0) | 1.2 (10.3) | -16.7 (19.9) | 0.5 (11.2)
  Global health status/QoL: Change at Cycle 2 Day 1: number analyzed (Participants) | 127 | 142 | 82 | 84
  Global health status/QoL: Change at Cycle 2 Day 1 | -9.8 (19.7) | -1.2 (14.5) | -10.9 (17.6) | 1.0 (10.8)
  Global health status/QoL: Change at Cycle 2 Day 15: number analyzed (Participants) | 118 | 134 | 80 | 80
  Global health status/QoL: Change at Cycle 2 Day 15 | -11.5 (21.0) | 0.2 (13.5) | -9.5 (18.0) | -1.4 (14.4)
  Global health status/QoL: Change at Cycle 3 Day 1: number analyzed (Participants) | 119 | 129 | 81 | 78
  Global health status/QoL: Change at Cycle 3 Day 1 | -10.6 (19.0) | -1.0 (14.6) | -9.4 (17.0) | -0.9 (14.6)
  Global health status/QoL: Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 129 | 78 | 76
  Global health status/QoL: Change at Cycle 4 Day 1 | -10.2 (19.6) | -1.0 (14.9) | -8.4 (18.9) | -1.8 (15.4)
  Global health status/QoL: Change at Cycle 5 Day 1: number analyzed (Participants) | 110 | 116 | 72 | 64
  Global health status/QoL: Change at Cycle 5 Day 1 | -12.0 (20.4) | -0.1 (15.1) | -8.9 (17.3) | 0.4 (16.6)
  Global health status/QoL: Change at Cycle 6 Day 1: number analyzed (Participants) | 106 | 112 | 69 | 63
  Global health status/QoL: Change at Cycle 6 Day 1 | -8.9 (18.9) | -2.2 (16.1) | -12.4 (19.3) | -0.5 (16.5)
  Global health status/QoL: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 108 | 68 | 59
  Global health status/QoL: Change at Cycle 7 Day 1 | -10.7 (19.4) | -1.6 (16.8) | -11.8 (17.9) | -2.3 (15.8)
  Global health status/QoL: Change at Cycle 8 Day 1: number analyzed (Participants) | 104 | 106 | 65 | 53
  Global health status/QoL: Change at Cycle 8 Day 1 | -10.3 (18.3) | -1.6 (17.6) | -11.2 (20.5) | -3.3 (17.0)
  Global health status/QoL: Change at Cycle 9 Day 1: number analyzed (Participants) | 100 | 101 | 63 | 52
  Global health status/QoL: Change at Cycle 9 Day 1 | -11.3 (21.9) | -0.5 (16.9) | -8.3 (19.7) | -1.6 (16.6)
  Global health status/QoL: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 63 | 47
  Global health status/QoL: Change at Cycle 10 Day 1 | -7.6 (19.1) | -0.7 (15.9) | -9.8 (18.7) | 0.2 (15.0)
  Global health status/QoL: Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 93 | 57 | 48
  Global health status/QoL: Change at Cycle 11 Day 1 | -7.8 (19.5) | -0.8 (15.3) | -8.8 (18.9) | -3.1 (18.2)
  Global health status/QoL: Change at Cycle 12 Day 1: number analyzed (Participants) | 90 | 91 | 55 | 48
  Global health status/QoL: Change at Cycle 12 Day 1 | -9.3 (20.2) | -0.8 (16.0) | -10.5 (17.4) | -3.6 (18.0)
  Global health status/QoL: Change at Cycle 13 Day 1: number analyzed (Participants) | 82 | 89 | 54 | 45
  Global health status/QoL: Change at Cycle 13 Day 1 | -7.5 (17.5) | -3.4 (19.4) | -9.4 (18.9) | -3.9 (15.8)
  Global health status/QoL: Change at EOT: number analyzed (Participants) | 123 | 125 | 67 | 75
  Global health status/QoL: Change at EOT | -5.2 (19.0) | -3.6 (19.0) | -3.0 (18.4) | -7.4 (21.7)
  Global health status/QoL: Change at PT 13 Weeks: number analyzed (Participants) | 90 | 74 | 56 | 38
  Global health status/QoL: Change at PT 13 Weeks | 0.1 (16.0) | -0.1 (15.7) | -1.0 (18.1) | 0.2 (20.0)
  Global health status/QoL: Change at PT 26 Weeks: number analyzed (Participants) | 90 | 72 | 47 | 35
  Global health status/QoL: Change at PT 26 Weeks | -2.2 (16.2) | 0.5 (14.8) | 0.4 (19.5) | 0.0 (19.7)
  Global health status/QoL: Change at PT 39 Weeks: number analyzed (Participants) | 79 | 68 | 41 | 33
  Global health status/QoL: Change at PT 39 Weeks | -4.1 (21.6) | -0.9 (15.2) | -0.4 (16.9) | -1.3 (19.9)
  Global health status/QoL: Change at PT 52 Weeks: number analyzed (Participants) | 76 | 62 | 27 | 25
  Global health status/QoL: Change at PT 52 Weeks | -2.3 (15.6) | -0.7 (15.3) | 2.2 (13.2) | -2.0 (23.6)
  Global health status/QoL: Change at PT 65 Weeks: number analyzed (Participants) | 53 | 38 | 17 | 18
  Global health status/QoL: Change at PT 65 Weeks | -0.9 (17.7) | -2.0 (15.1) | 1.5 (15.1) | -0.5 (17.7)
  Global health status/QoL: Change at PT 78 Weeks: number analyzed (Participants) | 46 | 33 | 15 | 9
  Global health status/QoL: Change at PT 78 Weeks | -0.9 (15.6) | -1.5 (15.8) | 1.7 (14.8) | -0.9 (13.5)
  Global health status/QoL: Change at PT 91 Weeks: number analyzed (Participants) | 33 | 29 | 15 | 12
  Global health status/QoL: Change at PT 91 Weeks | 0.3 (17.4) | -2.6 (17.6) | 6.1 (15.3) | -2.1 (24.7)
  Global health status/QoL: Change at PT 104 Weeks: number analyzed (Participants) | 27 | 25 | 10 | 9
  Global health status/QoL: Change at PT 104 Weeks | 1.2 (14.9) | -4.7 (19.4) | -3.3 (19.3) | 0.0 (29.2)
  Global health status/QoL: Change at PT 117 Weeks: number analyzed (Participants) | 22 | 17 | 8 | 5
  Global health status/QoL: Change at PT 117 Weeks | 0.4 (20.5) | 2.5 (15.0) | -1.0 (13.7) | 6.7 (21.6)
  Global health status/QoL: Change at PT 130 Weeks: number analyzed (Participants) | 16 | 12 | 5 | 5
  Global health status/QoL: Change at PT 130 Weeks | 2.1 (7.1) | -3.5 (16.8) | -3.3 (12.6) | 5.0 (24.0)
  Global health status/QoL: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Global health status/QoL: Change at PT 143 Weeks | -1.2 (18.9) | -4.2 (5.9) | -11.1 (9.6) | -8.3 (11.8)
  Global health status/QoL: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Global health status/QoL: Change at PT 156 Weeks | 11.1 (4.8) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable |  | 12.5 (5.9)
  Global health status/QoL: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Global health status/QoL: Change at PT 169 Weeks | 8.3 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Global health status/QoL: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Global health status/QoL: Change at PT 182 Weeks | 19.4 (12.7) |  |  |
  Global health status/QoL: Change at PT/Discontin.: number analyzed (Participants) | 8 | 1 | 6 | 1
  Global health status/QoL: Change at PT/Discontin. | -4.2 (19.9) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. | 0.0 (31.2) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable.
  Role functioning: Cycle 1 Day 1 (Baseline) | 86.7 (21.9) | 87.2 (22.5) | 86.6 (22.0) | 88.6 (23.2)
  Role functioning: Change at Cycle 1 Day 8: number analyzed (Participants) | 24 | 22 | 16 | 19
  Role functioning: Change at Cycle 1 Day 8 | -2.8 (15.3) | -0.8 (10.9) | -1.0 (16.6) | 4.4 (18.3)
  Role functioning: Change at Cycle 1 Day 15: number analyzed (Participants) | 132 | 139 | 80 | 84
  Role functioning: Change at Cycle 1 Day 15 | -19.4 (29.1) | 0.2 (16.3) | -15.2 (27.6) | -2.4 (19.6)
  Role functioning: Change at Cycle 1 Day 22: number analyzed (Participants) | 22 | 21 | 15 | 17
  Role functioning: Change at Cycle 1 Day 22 | -10.6 (28.4) | 1.6 (9.0) | -16.7 (20.9) | -1.0 (25.3)
  Role functioning: Change at Cycle 2 Day 1: number analyzed (Participants) | 127 | 142 | 83 | 84
  Role functioning: Change at Cycle 2 Day 1 | -13.0 (26.6) | 0.2 (16.6) | -13.3 (27.5) | 0.4 (17.5)
  Role functioning: Change at Cycle 2 Day 15: number analyzed (Participants) | 119 | 134 | 80 | 81
  Role functioning: Change at Cycle 2 Day 15 | -11.1 (25.7) | -0.6 (18.4) | -9.6 (21.5) | -0.4 (17.5)
  Role functioning: Change at Cycle 3 Day 1: number analyzed (Participants) | 119 | 129 | 81 | 78
  Role functioning: Change at Cycle 3 Day 1 | -9.7 (25.4) | 0.4 (19.0) | -8.2 (21.3) | -2.1 (21.2)
  Role functioning: Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 129 | 78 | 76
  Role functioning: Change at Cycle 4 Day 1 | -8.4 (23.8) | 0.3 (21.3) | -9.0 (19.7) | -1.3 (19.0)
  Role functioning: Change at Cycle 5 Day 1: number analyzed (Participants) | 110 | 117 | 72 | 64
  Role functioning: Change at Cycle 5 Day 1 | -11.1 (26.0) | 0.6 (20.5) | -10.4 (22.3) | 0.8 (22.7)
  Role functioning: Change at Cycle 6 Day 1: number analyzed (Participants) | 106 | 111 | 69 | 63
  Role functioning: Change at Cycle 6 Day 1 | -5.8 (24.2) | -0.5 (18.3) | -11.6 (22.9) | 0.5 (20.1)
  Role functioning: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 108 | 68 | 59
  Role functioning: Change at Cycle 7 Day 1 | -9.9 (27.6) | 0.9 (21.5) | -8.8 (24.0) | 0.3 (21.3)
  Role functioning: Change at Cycle 8 Day 1: number analyzed (Participants) | 105 | 105 | 65 | 53
  Role functioning: Change at Cycle 8 Day 1 | -9.2 (26.5) | -1.9 (23.0) | -9.5 (24.5) | -0.3 (21.3)
  Role functioning: Change at Cycle 9 Day 1: number analyzed (Participants) | 100 | 100 | 63 | 52
  Role functioning: Change at Cycle 9 Day 1 | -11.2 (28.4) | 0.0 (20.7) | -7.9 (23.5) | -1.9 (25.7)
  Role functioning: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 63 | 47
  Role functioning: Change at Cycle 10 Day 1 | -8.5 (25.5) | -1.7 (19.3) | -7.7 (23.2) | 3.9 (22.3)
  Role functioning: Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 93 | 57 | 48
  Role functioning: Change at Cycle 11 Day 1 | -6.6 (24.5) | -1.3 (19.7) | -10.2 (25.0) | -3.5 (24.8)
  Role functioning: Change at Cycle 12 Day 1: number analyzed (Participants) | 90 | 91 | 55 | 48
  Role functioning: Change at Cycle 12 Day 1 | -8.7 (26.2) | -0.4 (17.2) | -8.2 (25.2) | 0.3 (26.3)
  Role functioning: Change at Cycle 13 Day 1: number analyzed (Participants) | 82 | 89 | 54 | 45
  Role functioning: Change at Cycle 13 Day 1 | -8.1 (24.6) | -4.5 (22.2) | -8.3 (25.9) | -2.2 (24.3)
  Role functioning: Change at End Of Treatment: number analyzed (Participants) | 123 | 125 | 67 | 75
  Role functioning: Change at End Of Treatment | -4.7 (25.0) | -1.3 (23.2) | -4.2 (25.0) | -6.0 (27.6)
  Role functioning: Change at PT 13 Weeks: number analyzed (Participants) | 90 | 74 | 56 | 38
  Role functioning: Change at PT 13 Weeks | 2.0 (21.8) | 1.8 (17.6) | 1.2 (19.0) | 5.3 (26.9)
  Role functioning: Change at PT 26 Weeks: number analyzed (Participants) | 90 | 72 | 47 | 35
  Role functioning: Change at PT 26 Weeks | 0.9 (24.7) | 3.0 (17.3) | 0.4 (20.1) | 5.2 (24.5)
  Role functioning: Change at PT 39 Weeks: number analyzed (Participants) | 79 | 68 | 42 | 33
  Role functioning: Change at PT 39 Weeks | 2.7 (24.2) | 0.2 (21.1) | 0.4 (21.3) | 7.1 (28.0)
  Role functioning: Change at PT 52 Weeks: number analyzed (Participants) | 76 | 62 | 27 | 25
  Role functioning: Change at PT 52 Weeks | 2.4 (23.8) | 0.8 (20.3) | 0.6 (18.2) | 4.0 (29.0)
  Role functioning: Change at PT 65 Weeks: number analyzed (Participants) | 53 | 38 | 17 | 18
  Role functioning: Change at PT 65 Weeks | 5.3 (19.3) | -1.3 (16.6) | 3.9 (11.1) | 7.4 (29.3)
  Role functioning: Change at PT 78 Weeks: number analyzed (Participants) | 46 | 33 | 15 | 9
  Role functioning: Change at PT 78 Weeks | -1.4 (25.5) | -4.0 (20.0) | 4.4 (11.7) | -3.7 (13.9)
  Role functioning: Change at PT 91 Weeks: number analyzed (Participants) | 33 | 29 | 15 | 12
  Role functioning: Change at PT 91 Weeks | 3.5 (27.2) | -1.7 (17.4) | 1.1 (14.7) | 16.7 (35.5)
  Role functioning: Change at PT 104 Weeks: number analyzed (Participants) | 27 | 25 | 10 | 9
  Role functioning: Change at PT 104 Weeks | 6.2 (22.2) | -7.3 (20.5) | 6.7 (14.1) | 14.8 (38.6)
  Role functioning: Change at PT 117 Weeks: number analyzed (Participants) | 22 | 17 | 9 | 5
  Role functioning: Change at PT 117 Weeks | 7.6 (26.6) | -2.0 (10.0) | 5.6 (11.8) | 26.7 (41.8)
  Role functioning: Change at PT 130 Weeks: number analyzed (Participants) | 17 | 12 | 5 | 5
  Role functioning: Change at PT 130 Weeks | 6.9 (21.3) | -5.6 (14.8) | 3.3 (18.3) | 23.3 (43.5)
  Role functioning: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Role functioning: Change at PT 143 Weeks | 7.1 (18.9) | 0.0 (0.0) | 11.1 (19.2) | 8.3 (11.8)
  Role functioning: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Role functioning: Change at PT 156 Weeks | 27.8 (25.5) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  | 16.7 (23.6)
  Role functioning: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Role functioning: Change at PT 169 Weeks | 16.7 (23.6) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Role functioning: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Role functioning: Change at PT 182 Weeks | 27.8 (25.5) |  |  |
  Role functioning: Change at PT/Discontin.: number analyzed (Participants) | 8 | 1 | 6 | 1
  Role functioning: Change at PT/Discontin. | -8.3 (23.6) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. | 11.1 (17.2) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable.
  Social functioning: Cycle 1 Day 1 (Baseline) | 89.6 (16.6) | 88.2 (20.8) | 87.7 (21.2) | 90.4 (19.9)
  Social functioning: Change at Cycle 1 Day 8: number analyzed (Participants) | 24 | 22 | 16 | 19
  Social functioning: Change at Cycle 1 Day 8 | 1.4 (18.3) | 0.8 (12.0) | 2.1 (14.8) | 0.9 (8.7)
  Social functioning: Change at Cycle 1 Day 15: number analyzed (Participants) | 132 | 139 | 78 | 84
  Social functioning: Change at Cycle 1 Day 15 | -15.0 (26.9) | 0.8 (13.8) | -7.5 (18.9) | 0.4 (13.4)
  Social functioning: Change at Cycle 1 Day 22: number analyzed (Participants) | 22 | 21 | 15 | 17
  Social functioning: Change at Cycle 1 Day 22 | -9.1 (28.0) | 5.6 (13.3) | -5.6 (17.4) | -2.0 (20.3)
  Social functioning: Change at Cycle 2 Day 1: number analyzed (Participants) | 127 | 142 | 82 | 84
  Social functioning: Change at Cycle 2 Day 1 | -8.0 (22.9) | 2.2 (16.6) | -10.2 (23.8) | 3.0 (13.7)
  Social functioning: Change at Cycle 2 Day 15: number analyzed (Participants) | 118 | 134 | 80 | 80
  Social functioning: Change at Cycle 2 Day 15 | -8.3 (21.5) | 2.7 (16.9) | -7.7 (18.2) | 4.0 (17.0)
  Social functioning: Change at Cycle 3 Day 1: number analyzed (Participants) | 119 | 129 | 81 | 78
  Social functioning: Change at Cycle 3 Day 1 | -8.1 (21.5) | 2.3 (17.8) | -7.4 (21.1) | 1.5 (17.9)
  Social functioning: Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 129 | 78 | 76
  Social functioning: Change at Cycle 4 Day 1 | -7.1 (21.5) | 1.7 (18.1) | -7.5 (20.6) | 1.3 (13.5)
  Social functioning: Change at Cycle 5 Day 1: number analyzed (Participants) | 110 | 116 | 72 | 64
  Social functioning: Change at Cycle 5 Day 1 | -9.4 (21.7) | 3.3 (17.6) | -9.5 (18.5) | 2.6 (18.6)
  Social functioning: Change at Cycle 6 Day 1: number analyzed (Participants) | 106 | 112 | 69 | 63
  Social functioning: Change at Cycle 6 Day 1 | -7.2 (22.2) | 1.9 (17.6) | -11.4 (22.4) | 0.0 (17.2)
  Social functioning: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 108 | 68 | 59
  Social functioning: Change at Cycle 7 Day 1 | -8.0 (22.7) | 4.5 (17.0) | -9.6 (22.9) | 0.0 (17.2)
  Social functioning: Change at Cycle 8 Day 1: number analyzed (Participants) | 104 | 106 | 65 | 53
  Social functioning: Change at Cycle 8 Day 1 | -8.3 (23.6) | 2.2 (17.7) | -7.9 (23.0) | 0.6 (16.0)
  Social functioning: Change at Cycle 9 Day 1: number analyzed (Participants) | 100 | 101 | 63 | 52
  Social functioning: Change at Cycle 9 Day 1 | -11.0 (26.2) | 1.7 (19.7) | -8.2 (22.8) | -3.8 (21.5)
  Social functioning: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 63 | 47
  Social functioning: Change at Cycle 10 Day 1 | -8.7 (24.9) | 0.0 (16.1) | -8.7 (23.4) | -0.7 (16.3)
  Social functioning: Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 93 | 57 | 48
  Social functioning: Change at Cycle 11 Day 1 | -8.6 (24.4) | 1.4 (15.1) | -9.9 (23.1) | -2.1 (21.6)
  Social functioning: Change at Cycle 12 Day 1: number analyzed (Participants) | 90 | 91 | 55 | 48
  Social functioning: Change at Cycle 12 Day 1 | -10.6 (24.2) | -0.4 (15.7) | -9.1 (22.2) | 0.0 (16.5)
  Social functioning: Change at Cycle 13 Day 1: number analyzed (Participants) | 82 | 89 | 54 | 45
  Social functioning: Change at Cycle 13 Day 1 | -8.3 (24.2) | -1.9 (21.1) | -10.2 (25.2) | 1.5 (17.7)
  Social functioning: Change at End of Treatment: number analyzed (Participants) | 123 | 125 | 67 | 75
  Social functioning: Change at End of Treatment | -6.1 (21.8) | 1.2 (25.8) | -5.5 (23.3) | -3.3 (21.2)
  Social functioning: Change at PT 13 Weeks: number analyzed (Participants) | 90 | 74 | 56 | 38
  Social functioning: Change at PT 13 Weeks | -1.7 (18.9) | 2.7 (15.4) | 1.2 (16.2) | 1.3 (19.5)
  Social functioning: Change at PT 26 Weeks: number analyzed (Participants) | 90 | 72 | 47 | 35
  Social functioning: Change at PT 26 Weeks | -2.6 (20.3) | 4.2 (15.0) | 0.0 (13.9) | 2.4 (14.1)
  Social functioning: Change at PT 39 Weeks: number analyzed (Participants) | 79 | 68 | 41 | 33
  Social functioning: Change at PT 39 Weeks | 3.4 (16.5) | 2.7 (15.4) | 0.0 (18.3) | 5.1 (17.4)
  Social functioning: Change at PT 52 Weeks: number analyzed (Participants) | 76 | 62 | 27 | 25
  Social functioning: Change at PT 52 Weeks | -0.7 (18.9) | 1.6 (14.7) | 2.5 (13.6) | -1.3 (18.0)
  Social functioning: Change at PT 65 Weeks: number analyzed (Participants) | 53 | 38 | 17 | 18
  Social functioning: Change at PT 65 Weeks | 2.8 (18.7) | 0.9 (16.0) | 4.9 (11.4) | 0.9 (10.7)
  Social functioning: Change at PT 78 Weeks: number analyzed (Participants) | 46 | 33 | 15 | 9
  Social functioning: Change at PT 78 Weeks | 0.7 (20.8) | 6.1 (14.3) | 4.4 (13.3) | -1.9 (13.0)
  Social functioning: Change at PT 91 Weeks: number analyzed (Participants) | 32 | 29 | 15 | 12
  Social functioning: Change at PT 91 Weeks | 2.6 (21.6) | 1.7 (20.1) | 2.2 (13.9) | 2.8 (12.0)
  Social functioning: Change at PT 104 Weeks: number analyzed (Participants) | 27 | 25 | 10 | 9
  Social functioning: Change at PT 104 Weeks | 2.5 (18.3) | 0.0 (19.2) | 3.3 (10.5) | 1.9 (13.0)
  Social functioning: Change at PT 117 Weeks: number analyzed (Participants) | 22 | 17 | 8 | 5
  Social functioning: Change at PT 117 Weeks | 9.1 (15.2) | 2.0 (21.1) | -2.1 (5.9) | 3.3 (18.3)
  Social functioning: Change at PT 130 Weeks: number analyzed (Participants) | 17 | 12 | 5 | 5
  Social functioning: Change at PT 130 Weeks | 9.8 (15.7) | 6.9 (16.6) | 0.0 (0.0) | 10.0 (32.5)
  Social functioning: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Social functioning: Change at PT 143 Weeks | 7.1 (18.9) | 0.0 (0.0) | 0.0 (0.0) | -8.3 (11.8)
  Social functioning: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Social functioning: Change at PT 156 Weeks | 27.8 (9.6) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  | 0.0 (0.0)
  Social functioning: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Social functioning: Change at PT 169 Weeks | 25.0 (11.8) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Social functioning: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Social functioning: Change at PT 182 Weeks | 27.8 (9.6) |  |  |
  Social functioning: Change at PT/Discontinuation: number analyzed (Participants) | 8 | 1 | 6 | 1
  Social functioning: Change at PT/Discontinuation | -4.2 (21.4) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. | 0.0 (10.5) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable.
  Insomnia: Cycle 1 Day 1 (Baseline) | 18.4 (23.2) | 17.0 (25.4) | 17.2 (23.2) | 18.7 (24.6)
  Insomnia: Change at Cycle 1 Day 8: number analyzed (Participants) | 24 | 22 | 16 | 19
  Insomnia: Change at Cycle 1 Day 8 | 11.1 (18.8) | -3.0 (14.2) | 2.1 (22.7) | 1.8 (20.7)
  Insomnia: Change at Cycle 1 Day 15: number analyzed (Participants) | 132 | 139 | 80 | 84
  Insomnia: Change at Cycle 1 Day 15 | 6.8 (29.6) | 1.0 (19.6) | 9.6 (26.1) | -4.4 (21.2)
  Insomnia: Change at Cycle 1 Day 22: number analyzed (Participants) | 22 | 21 | 15 | 17
  Insomnia: Change at Cycle 1 Day 22 | 9.1 (27.6) | -3.2 (23.3) | 6.7 (18.7) | -7.8 (22.1)
  Insomnia: Change at Cycle 2 Day 1: number analyzed (Participants) | 127 | 142 | 83 | 84
  Insomnia: Change at Cycle 2 Day 1 | 0.8 (23.9) | -1.2 (22.6) | 2.4 (24.8) | -5.6 (19.9)
  Insomnia: Change at Cycle 2 Day 15: number analyzed (Participants) | 119 | 134 | 80 | 81
  Insomnia: Change at Cycle 2 Day 15 | 5.9 (27.7) | 0.5 (25.2) | 2.1 (28.7) | -3.7 (23.0)
  Insomnia: Change at Cycle 3 Day 1: number analyzed (Participants) | 119 | 129 | 81 | 78
  Insomnia: Change at Cycle 3 Day 1 | 0.6 (25.7) | -1.3 (23.0) | -0.4 (28.1) | -2.6 (22.0)
  Insomnia: Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 129 | 78 | 75
  Insomnia: Change at Cycle 4 Day 1 | 2.2 (25.6) | -1.0 (25.0) | 3.4 (26.1) | -4.9 (23.1)
  Insomnia: Change at Cycle 5 Day 1: number analyzed (Participants) | 110 | 117 | 72 | 64
  Insomnia: Change at Cycle 5 Day 1 | 2.4 (27.4) | 0.3 (23.8) | 3.2 (26.9) | -5.7 (22.7)
  Insomnia: Change at Cycle 6 Day 1: number analyzed (Participants) | 106 | 112 | 68 | 63
  Insomnia: Change at Cycle 6 Day 1 | 3.1 (28.6) | 1.8 (25.6) | 3.4 (26.5) | -4.2 (24.3)
  Insomnia: Change at Cycle 7 Day 1: number analyzed (Participants) | 106 | 108 | 68 | 59
  Insomnia: Change at Cycle 7 Day 1 | 4.7 (26.6) | -0.3 (25.6) | 3.4 (23.8) | -2.3 (17.4)
  Insomnia: Change at Cycle 8 Day 1: number analyzed (Participants) | 104 | 106 | 65 | 53
  Insomnia: Change at Cycle 8 Day 1 | 4.2 (28.5) | 0.6 (29.1) | 7.7 (29.9) | -6.3 (18.6)
  Insomnia: Change at Cycle 9 Day 1: number analyzed (Participants) | 100 | 101 | 63 | 52
  Insomnia: Change at Cycle 9 Day 1 | 3.3 (27.8) | 0.7 (27.1) | 6.3 (28.6) | 0.0 (21.9)
  Insomnia: Change at Cycle 10 Day 1: number analyzed (Participants) | 96 | 97 | 63 | 47
  Insomnia: Change at Cycle 10 Day 1 | 1.7 (22.9) | 0.7 (22.0) | 4.2 (27.1) | -1.4 (19.6)
  Insomnia: Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 93 | 57 | 48
  Insomnia: Change at Cycle 11 Day 1 | 0.7 (25.0) | -0.7 (25.5) | 5.3 (32.0) | 1.4 (18.1)
  Insomnia: Change at Cycle 12 Day 1: number analyzed (Participants) | 89 | 91 | 55 | 48
  Insomnia: Change at Cycle 12 Day 1 | 0.7 (24.6) | 0.0 (27.7) | 3.6 (29.2) | 0.0 (23.8)
  Insomnia: Change at Cycle 13 Day 1: number analyzed (Participants) | 82 | 88 | 54 | 45
  Insomnia: Change at Cycle 13 Day 1 | 4.1 (26.4) | 3.8 (31.7) | 6.2 (29.0) | -1.5 (22.4)
  Insomnia: Change at End Of Treatment: number analyzed (Participants) | 123 | 125 | 67 | 75
  Insomnia: Change at End Of Treatment | -3.0 (25.3) | 1.3 (28.8) | 3.5 (32.4) | 0.4 (26.6)
  Insomnia: Change at PT 13 Weeks: number analyzed (Participants) | 90 | 74 | 56 | 38
  Insomnia: Change at PT 13 Weeks | -4.4 (21.9) | -1.8 (25.2) | -2.4 (24.5) | -0.9 (22.6)
  Insomnia: Change at PT 26 Weeks: number analyzed (Participants) | 90 | 72 | 47 | 35
  Insomnia: Change at PT 26 Weeks | -2.6 (21.9) | 0.5 (28.2) | -1.4 (23.0) | -3.8 (22.5)
  Insomnia: Change at PT 39 Weeks: number analyzed (Participants) | 79 | 68 | 42 | 33
  Insomnia: Change at PT 39 Weeks | -5.9 (23.7) | -0.5 (29.6) | -2.4 (27.9) | -5.1 (23.7)
  Insomnia: Change at PT 52 Weeks: number analyzed (Participants) | 76 | 62 | 27 | 25
  Insomnia: Change at PT 52 Weeks | -3.9 (24.3) | 0.5 (26.6) | -2.5 (26.0) | -8.0 (26.0)
  Insomnia: Change at PT 65 Weeks: number analyzed (Participants) | 53 | 38 | 17 | 18
  Insomnia: Change at PT 65 Weeks | -6.3 (23.6) | 1.8 (21.8) | -3.9 (33.1) | -3.7 (22.5)
  Insomnia: Change at PT 78 Weeks: number analyzed (Participants) | 46 | 33 | 15 | 9
  Insomnia: Change at PT 78 Weeks | -2.2 (28.5) | 1.0 (30.6) | -4.4 (27.8) | -3.7 (26.1)
  Insomnia: Change at PT 91 Weeks: number analyzed (Participants) | 33 | 29 | 15 | 12
  Insomnia: Change at PT 91 Weeks | -4.0 (16.2) | -1.1 (25.9) | -4.4 (21.3) | -2.8 (26.4)
  Insomnia: Change at PT 104 Weeks: number analyzed (Participants) | 27 | 25 | 10 | 9
  Insomnia: Change at PT 104 Weeks | -4.9 (17.8) | 4.0 (27.8) | 0.0 (22.2) | -3.7 (11.1)
  Insomnia: Change at PT 117 Weeks: number analyzed (Participants) | 22 | 17 | 9 | 5
  Insomnia: Change at PT 117 Weeks | -9.1 (18.3) | -7.8 (30.1) | 0.0 (16.7) | -13.3 (29.8)
  Insomnia: Change at PT 130 Weeks: number analyzed (Participants) | 17 | 12 | 5 | 5
  Insomnia: Change at PT 130 Weeks | -7.8 (22.1) | -8.3 (20.7) | 6.7 (27.9) | -6.7 (14.9)
  Insomnia: Change at PT 143 Weeks: number analyzed (Participants) | 7 | 2 | 3 | 2
  Insomnia: Change at PT 143 Weeks | -14.3 (17.8) | -16.7 (23.6) | 0.0 (33.3) | 0.0 (0.0)
  Insomnia: Change at PT 156 Weeks: number analyzed (Participants) | 3 | 1 | 0 | 2
  Insomnia: Change at PT 156 Weeks | -11.1 (19.2) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  | 0.0 (0.0)
  Insomnia: Change at PT 169 Weeks: number analyzed (Participants) | 2 | 1 | 0 | 0
  Insomnia: Change at PT 169 Weeks | 0.0 (0.0) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. |  |
  Insomnia: Change at PT 182 Weeks: number analyzed (Participants) | 3 | 0 | 0 | 0
  Insomnia: Change at PT 182 Weeks | -11.1 (19.2) |  |  |
  Insomnia: Change at PT/Discont.: number analyzed (Participants) | 8 | 1 | 6 | 1
  Insomnia: Change at PT/Discont. | 0.0 (17.8) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable. | 5.6 (25.1) | 0.0 (NA) — 1 participant was analyzed, so standard deviation is not applicable.

6. Secondary Outcome: Plasma Concentration of Vemurafenib
Time Frame: Pre-morning dose (0 hour [hr]) and 1 to 4 hrs post-dose on Days 1, 8, 15, and 22 of Cycle 1; pre-morning dose (0 hr) on Days 1 and 15 of Cycle 2; pre-morning dose (0 hr) on Day 1 of Cycles 3-13; at end of treatment (up to 13 months)
Population: The pharmacokinetic (PK)-evaluable population included all participants who received at least one dose of vemurafenib and had provided valid PK assessments.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort 1 Vemurafenib | Cohort 2 Vemurafenib
Number analyzed (Participants) | 149 | 92
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1 (nominal Day 1): number analyzed (Participants) | 122 | 77
  Cycle 1 Day 1 (nominal Day 1) | 2880 (2770) | 3050 (3010)
  Cycle 1 Day 8: number analyzed (Participants) | 79 | 52
  Cycle 1 Day 8 | 49900 (19800) | 43400 (13600)
  Cycle 1 Day 15: number analyzed (Participants) | 55 | 43
  Cycle 1 Day 15 | 45300 (23000) | 50200 (20500)
  Cycle 1 Day 22: number analyzed (Participants) | 49 | 45
  Cycle 1 Day 22 | 44000 (22400) | 48800 (23700)
  Cycle 2 Day 1: number analyzed (Participants) | 107 | 69
  Cycle 2 Day 1 | 40200 (24100) | 43800 (19400)
  Cycle 2 Day 15: number analyzed (Participants) | 102 | 68
  Cycle 2 Day 15 | 42400 (21700) | 44200 (21200)
  Cycle 3 Day 1: number analyzed (Participants) | 100 | 69
  Cycle 3 Day 1 | 46700 (21500) | 43700 (22000)
  Cycle 4 Day 1: number analyzed (Participants) | 98 | 68
  Cycle 4 Day 1 | 44800 (19300) | 47400 (20100)
  Cycle 5 Day 1: number analyzed (Participants) | 92 | 61
  Cycle 5 Day 1 | 43100 (18800) | 43700 (19400)
  Cycle 6 Day 1: number analyzed (Participants) | 82 | 62
  Cycle 6 Day 1 | 46000 (18900) | 42000 (22000)
  Cycle 7 Day 1: number analyzed (Participants) | 86 | 57
  Cycle 7 Day 1 | 42800 (20500) | 45200 (20500)
  Cycle 8 Day 1: number analyzed (Participants) | 81 | 55
  Cycle 8 Day 1 | 43600 (19900) | 42600 (18900)
  Cycle 9 Day 1: number analyzed (Participants) | 77 | 51
  Cycle 9 Day 1 | 42900 (18400) | 43000 (17700)
  Cycle 10 Day 1: number analyzed (Participants) | 38 | 29
  Cycle 10 Day 1 | 41000 (19000) | 43900 (18500)
  Cycle 11 Day 1: number analyzed (Participants) | 35 | 35
  Cycle 11 Day 1 | 45900 (15300) | 39700 (17600)
  Cycle 12 Day 1: number analyzed (Participants) | 34 | 26
  Cycle 12 Day 1 | 43700 (15200) | 46600 (19800)
  Cycle 13 Day 1: number analyzed (Participants) | 36 | 26
  Cycle 13 Day 1 | 44000 (17200) | 42600 (19900)

ADVERSE EVENTS:
Time Frame: Up to the data cutoff of July 13, 2018 (approximately 6 years).
Description: The safety population included all participants who received at least one dose of study medication.
Arm/Group | Cohort 1 Vemurafenib | Cohort 1 Placebo | Cohort 2 Vemurafenib | Cohort 2 Placebo
All-Cause Mortality (participants affected / at risk) | 18/154 | 33/156 | 25/93 | 26/91
Serious Adverse Events (participants affected / at risk) | 25/154 | 16/156 | 15/93 | 9/91
Other Adverse Events (participants affected / at risk) | 150/154 | 117/156 | 92/93 | 67/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Vemurafenib (N=154) | Cohort 1 Placebo (N=156) | Cohort 2 Vemurafenib (N=93) | Cohort 2 Placebo (N=91)
Pericarditis (Cardiac disorders) | 1 | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Leukoplakia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 1
Groin infection (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 7 | 3 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Vemurafenib (N=154) | Cohort 1 Placebo (N=156) | Cohort 2 Vemurafenib (N=93) | Cohort 2 Placebo (N=91)
Rash (Skin and subcutaneous tissue disorders) | 57 | 20 | 34 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 57 | 10 | 37 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 44 | 27 | 28 | 3
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 52 | 6 | 35 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 58 | 5 | 25 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 32 | 13 | 16 | 5
Erythema (Skin and subcutaneous tissue disorders) | 20 | 8 | 17 | 6
Actinic keratosis (Skin and subcutaneous tissue disorders) | 15 | 8 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 101 | 37 | 49 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 | 15 | 17 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 10 | 9 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 8 | 7 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 14 | 7 | 2
Fatigue (General disorders) | 52 | 52 | 26 | 18
Asthenia (General disorders) | 24 | 13 | 17 | 10
Pyrexia (General disorders) | 28 | 11 | 16 | 7
Oedema peripheral (General disorders) | 9 | 8 | 7 | 4
Nausea (Gastrointestinal disorders) | 59 | 36 | 27 | 9
Diarrhoea (Gastrointestinal disorders) | 38 | 32 | 27 | 9
Vomiting (Gastrointestinal disorders) | 19 | 9 | 14 | 4
Constipation (Gastrointestinal disorders) | 8 | 11 | 9 | 3
Abdominal pain (Gastrointestinal disorders) | 10 | 7 | 6 | 2
Headache (Nervous system disorders) | 29 | 32 | 20 | 11
Dysgeusia (Nervous system disorders) | 17 | 4 | 8 | 3
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 | 2 | 19 | 2
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 7 | 10 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 0 | 10 | 2
Alanine aminotransferase increased (Investigations) | 28 | 5 | 14 | 4
Aspartate aminotransferase increased (Investigations) | 18 | 5 | 11 | 3
Sunburn (Injury, poisoning and procedural complications) | 25 | 2 | 19 | 2
Decreased appetite (Metabolism and nutrition disorders) | 17 | 11 | 16 | 2
Insomnia (Psychiatric disorders) | 9 | 7 | 12 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 8 | 6 | 3
Nasopharyngitis (Infections and infestations) | 9 | 10 | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT01667419/Prot_001.pdf
  • Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT01667419/SAP_002.pdf